

# **Clinical Study Protocol**

PROTOCOL NUMBER
PP LNM 01

# **TITLE**

A Randomized, Prospective, Open Label, Multicenter Study Assessing the Safety and Utility of PINPOINT® Near Infrared Fluorescence Imaging in the Identification of Lymph Nodes in Subjects with Uterine and Cervical Malignancies who are Undergoing Lymph Node Mapping

SHORT TITLE FILM

**PROTOCOL VERSION** Version 6.0, August 25<sup>th</sup>, 2017

# **SPONSOR**

Novadaq Technologies Inc. 5090 Explorer Dr., Ste. 202, Mississauga, Ontario, Canada, L4W 4T9

## Confidential

This is a Novadaq Technologies Inc., document that contains confidential information. It is intended solely for the recipient clinical investigator(s) and must not be disclosed to any other party.

2017-08-25

#### PROTOCOL APPROVAL

**Protocol Number:** 

PP LNM 01

Title of Protocol:

A Randomized, Prospective, Open Label, Multicenter Study Assessing the Safety and Utility of PINPOINT® Near Infrared Fluorescence Imaging in the Identification of Lymph Nodes in Subjects with Uterine and Cervical

Malignancies who are Undergoing Lymph Node Mapping.

Version:

6.0, August 25th, 2017

Written by:

Jen Pendlebury on behalf of Yohan D'Souza, PhD Clinical

Regulatory Scientist Novadag

Technologies Inc.



## PROTOCOL APPROVAL

| Protocol Number: | PP LNM 01 |
|------------------|-----------|

Technologies Inc.

Title of Protocol: A Randomized, Prospective, Open Label, Multicenter Study Assessing the

Safety and Utility of PINPOINT® Near Infrared Fluorescence Imaging in the Identification of Lymph Nodes in Subjects with Uterine and Cervical

Malignancies who are Undergoing Lymph Node Mapping.

**Version:** 6.0, August 25<sup>th</sup>, 2017

| Approved by: | Cox Swaln | 08/25/2017 |
|---|---|---|
| | Lori Swalm<br>Sr. Vice President, Regulatory, | Date |
| | Clinical and Economic Affairs<br>Novadaq Technologies Inc. | |
| Approved by | | |
| Approved by: | | |
| | Matt McKittrick On behalf of Yohan D'Souza, PhD Clinical | Date |
| | Regulatory Scientist Novadaq | |



#### PROTOCOL APPROVAL

Protocol Number: PP LNM 01

Title of Protocol: A Randomized, Prospective, Open Label, Multicenter Study Assessing the

Safety and Utility of PINPOINT® Near Infrared Fluorescence Imaging in the Identification of Lymph Nodes in Subjects with Uterine and Cervical

Malignancies who are Undergoing Lymph Node Mapping.

**Version:** 6.0, August 25<sup>th</sup>, 2017

| Approved by | Ap | pro | ved | by |
|-------------|----|-----|-----|----|
|-------------|----|-----|-----|----|

Lori Swalm

Sr. Vice President, Regulatory, Clinical and Economic Affairs Novadaq Technologies Inc. Date

Approved by:

Matt McKittrick On behalf of

Yohan D'Souza, PhD Clinical Regulatory Scientist Novadaq

Technologies Inc.

8/25/17 **Date** 

## PROTOCOL APPROVAL

Protocol Number:

PP LNM 01

Title of Protocol: A Randomized, Prospective, Open Label, Multicenter Study Assessing the Safety and Utility of PINPOINT® Endoscopic Near Infrared Fluorescence Imaging in the Identification of Lymph Nodes in Subjects with Uterine and Cervical Malignancies who are Undergoing Lymph Node Mapping

Version:

6.0, August 25th, 2017

Approved by:

Michael Frumovitz, MD Study Principal Investigator

M.D. Anderson Cancer

Center

Date

3/27/17

Nadeem Abu-Rustum, MD Study Principal Investigator

Memorial Sloan Kettering

Cancer Center

Marie Plante, MD Study Principal Investigator

L'Hôtel-Dieu de Québec,

Date

Pedro Escobar, MD Study Principal Investigator

HIMA San Pablo

Date

Approved by:

Mark F. Munsell, MS Senior Research Statistician Department of Blostatistics M.D Anderson Cancer Center

Date

PINPOINT® for Lymph Node Mapping Clinical Study Protocol PP LNM 01



#### PROTOCOL APPROVAL

Protocol Number:

PP LNM 01

Title of Protocol: A Randomized, Prospective, Open Label, Multicenter Study Assessing the Safety and Utility of PINPOINT® Endoscopic Near Infrared Fluorescence Imaging in the Identification of Lymph Nodes in Subjects with Uterine and

Cervical Malignancies who are Undergoing Lymph Node Mapping

Version:

6.0, August 25th, 2017

Approved by:

Michael Frumovitz, MD Study Principal Investigator M.D. Anderson Cancer Center

Date

Nadeem Abu-Rustum, MD Study Principal Investigator

Memorial Sloan Kettering

Cancer Center

Date

Date

Marie Plante, MD Study Principal Investigator L'Hôtel-Dieu de Québec,

Date

Pedro Escobar, MD Study Principal Investigator HIMA San Pablo

Approved by:

Mark 7. Mansell 8/30/17 Mark F. Munsell, MS

Senior Research Statistician Department of Biostatistics M.D Anderson Cancer Center



#### PROTOCOL SUMMARY

#### Study Number and Title:

**PP LNM 01**: A Randomized, Prospective, Open Label Multicenter Study Assessing the Safety and Utility of PINPOINT® Endoscopic Fluorescence Imaging to Identify Lymph Nodes in Patients with Uterine and Cervical Malignancies who are Undergoing Lymph Node Mapping.

Clinical Phase: Pivotal / Investigational Device Study

## Study Objectives:

# Primary:

To assess the effectiveness of intraoperative PINPOINT Near-Infrared Fluorescence imaging in the identification of lymph nodes in subjects with uterine and cervical malignancies who are undergoing lymph node mapping.

#### Secondary:

- To evaluate the effectiveness of PINPOINT and Blue dye in the identification of at least one lymph node (confirmed to be lymphoid tissue) per subject.
- To assess the safety of interstitial injection of ICG for intraoperative lymphatic mapping.

## Study Design:

This is a randomized prospective, open label, multicenter study to assess the safety and effectiveness of PINPOINT® Near Infrared Fluorescence Imaging (PINPOINT) in identification of lymph nodes (LN) in subjects with uterine and cervical malignancies who are undergoing LN mapping. This is a non-inferiority within-patient comparison study to determine the effectiveness of PINPOINT in the identification of LNs compared to LNs identified with Blue dye (1% Isosulfan blue). Approximately 150 subjects will be enrolled at up to 10 centers in North America. Prior to enrolling study subjects, participating surgeons at each center will be trained to perform intraoperative identification and mapping of LNs with IC2000 and Blue dye. Participating surgeons will be required to have completed at least 10 LN mapping procedures with a minimum of 3 LN mapping cases performed with PINPOINT prior to the initiation of enrollment.

#### Screening:

Subjects diagnosed with International Federation of Gynecology and Obstetrics (FIGO) clinical stage I endometrial or cervical cancer scheduled for surgery that includes clinically indicated LN mapping will be evaluated at baseline to determine if they meet the inclusion/exclusion criteria of the protocol. Subjects will be assessed to determine overall health status including demographics, vital signs, diagnosis and relevant medical history/underlying conditions. Eligible subjects who provide informed consent will be considered for inclusion into the study.

#### Day 0:

On the day of surgery subjects will be randomized (1:1) to either the Blue-PINPOINT (B-P) Arm or the PINPOINT-BLUE (P-B) Arm. Subjects in each arm will be randomized according to an independently generated randomization scheme to undergo lymphatic mapping with Blue dye first followed by mapping with PINPOINT (B-P Arm) or to undergo lymphatic mapping with PINPOINT first followed by mapping with Blue dye (P-B Arm).

Minimally invasive surgery will be performed according to the surgeon's standard practice.

The cervix will be injected four (4) times with a 1 ml solution Blue dye (1% solution: 10mg/ml) for a total dose of 40 mg and four (4) times with 1 ml of a 1.25 mg/ml solution of IC2000 for a total dose of 5 mg. The injection of Blue dye and IC2000 will occur while the subject is under anesthesia in the operating room.



In order to minimize the spillage of Blue dye or IC2000 interfering with the mapping procedure when LNs are excised, mapping will be performed on one side of the pelvis followed by other side and mapping with both Blue dye and PINPOINT will be performed prior to the excision of any LNs.

Subjects randomized into the B-P Arm will be administered Blue dye first followed by the administration of IC2000 and undergo LN mapping with Blue dye first followed by mapping with PINPOINT. LN mapping with Blue dye will be performed until the investigator identifies all blue nodes or determines that blue nodes cannot be identified. Once complete, the Investigator will begin mapping with PINPOINT until all 'IC2000' nodes are identified or the investigator determines that 'IC2000' nodes cannot be identified. Once mapping with both Blue dye and PINPOINT have been completed and documented, all LNs identified with Blue dye or PINPOINT will be excised.

Subjects randomized into the P-B Arm will be administered IC2000 first followed by the administration of Blue dye and undergo LN mapping with PINPOINT first followed by mapping with Blue dye. LN mapping with PINPOINT will be performed until the investigator identifies all 'IC2000' nodes or determines that 'IC2000' nodes cannot be identified. Once complete, the Investigator will begin mapping with Blue dye until all 'blue' nodes are identified or the investigator determines that 'blue' nodes cannot be identified. Once mapping with both Blue dye and PINPOINT have been completed and documented, LNs identified with Blue dye or PINPOINT will be excised.

Bilateral LN mapping for Clinical Stage I endometrial cancer will be performed according to the *NCCN Guidelines for Uterine Neoplasms, SLN Algorithm for Surgical Staging of Endometrial Cancer;* and LN mapping for Clinical Stage I cervical cancer will be performed according to the *NCCN Guidelines for Cervical Neoplasms, Surgical/SLN Mapping Algorithm for Early-Stage Cervical Cancer*<sup>1,2</sup>.

The surgeon will identify LN and lymphatic vessels based on visualization with white light for blue dye or PINPOINT for IC2000.

## LN Mapping with PINPOINT:

Intraoperative identification of LNs with IC2000 will be based on the following criteria:

- Direct visual identification of a node by NIR fluorescence with IC2000 using PINPOINT.
- Visibly or palpably abnormal lymph nodes designated as palpable masses and excised regardless of visible fluorescence.

Mapping will be considered complete when all nodes meeting any of the criteria above are identified and documented and the surgeon has scanned the full 360-degree area within the abdominal cavity. Fluorescent ducts should be followed in both directions in order to identify LNs to be excised.

#### LN Mapping with Blue dye:

Intraoperative identification of LNs with Blue dye will be based on the following criteria:

- Direct visual identification of a node stained with Blue dye.
- Visibly or palpably abnormal lymph nodes designated as palpable masses and excised regardless of visible blue dye.

Mapping will be considered complete when all nodes meeting any of the criteria above are identified and documented and the surgeon has scanned the full 360-degree area within the abdominal cavity Blue ducts should be followed in both directions in order to identify LNs to be excised.

#### Classification of LNs:

All LNs identified will be classified as:

- 1. Fluorescent only
- 2. Blue only
- 3. Both (Fluorescent and blue)
- 4. Abnormal or palpably hard (non-stained)
- 5. Non-stained node found at origin or termination of fluorescent duct
- 6. Non-stained node found at origin or termination of blue duct



7. Non-stained node found at origin or termination of fluorescent and blue duct

Effectiveness of intraoperative Blue dye in identifying LNs will be based on the proportion of LNs identified by visualization under white light and confirmed as lymphoid tissue by histology divided by the total number of LNs identified and excised.

Effectiveness of intraoperative PINPOINT in identifying LNs will be based on the proportion of LNs identified by PINPOINT and confirmed as lymphoid tissue by histology divided by the total number of LNs identified and excised.

Details of the surgery, including intraoperative findings will be documented. Surgical data will be collected including the ability to identify LNs the number of LNs identified and removed, the ability to unilaterally and bilaterally map LNs, and the anatomical location and distribution of identified LNs. Failed mapping is defined as no LNs detected.

Follow-up and Post-operative Complications:

Subjects will have standard of care assessments throughout the study according to the hospital/institution's standard procedures as well as study specific visits to monitor occurrence of any adverse events/ adverse device effects on the date of discharge and Day 30 (±7 days).

# Study Population

To be eligible for the study, subjects must meet the following main inclusion criteria:

- · 18 years of age or older
- Subjects with FIGO Clinical Stage I endometrial cancer undergoing minimally invasive hysterectomy with lymph node mapping.
- Subjects with FIGO Clinical Stage IA cervical cancer ≤ 2 cm in size undergoing minimally invasive hysterectomy, trachelectomy, or conization with lymph node mapping. Subjects with clinical Stage IA1 cervical cancer without lympho vascular space involvement (LVSI) and negative margins on cone biopsy are not to be included.
- Subjects with negative nodal status (N0)
- Subjects with negative metastatic involvement (M0).

Subjects meeting any of the following criteria will be excluded from the study:

- · Have had prior dissection and/or radiation in pelvis.
- Advanced cervical or endometrial cancer, T3/T4 lesions
- Diagnosis of cervical cancer with a tumor size greater than 2 cm.
- Locally advanced or inflammatory cervical or uterine cancer
- · Metastatic cervical or uterine cancer.
- · Known allergy or history of adverse reaction to ICG, iodine or iodine dyes.
- Known allergy or history of adverse reaction to Blue dye (Isosulfan blue) or triphenylmethane.
- Hepatic dysfunction defined as MELD Score > 12.
- Renal dysfunction defined as serum creatinine ≥ 2.0 mg/dl.
- Subjects who have participated in another investigational study within 30 days prior to surgery.
- · Pregnant or lactating subjects.
- Subjects who, in the Investigator's opinion, have any medical condition that makes the subject a poor candidate for the investigational procedure, or interferes with the interpretation of study results.



## Study Devices and Imaging Agents:

PINPOINT® Endoscopic Fluorescence Imaging System

An endoscopic fluorescence imaging system for high definition (HD) visible (VIS) light and near infrared (NIR) fluorescence imaging that includes the following components:

- · A surgical endoscope optimized for VIS/NIR illumination and imaging.
- A camera head that is also optimized for VIS/NIR imaging and mounts to the endoscope eyepiece
- · A flexible light guide cable.
- An endoscopic Video Processor/Illuminator for VIS/NIR illumination to the surgical endoscope via a flexible light guide cable, and the image processing required to generate simultaneous, real-time HD video color and NIR fluorescence images.
- · A high-definition medical video recorder that allows the capture of still images and video.
- The PINPOINT kit containing the imaging agent and aqueous solvent.

The imaging agent used with PINPOINT is ICG, which is a sterile, water-soluble tricarbocyanine dye with a peak spectral absorption at 800-810 nm in blood plasma or blood. ICG contains not more than 5.0% sodium iodide. In this study, investigational ICG, IC2000, will be administered to subjects.

Isosufan Blue 1% (Mylan) is a water-soluble contrast dye and is administered as a 1% solution for the purposes of lymphography.

## Study Variables:

## **Primary Variables**

Effectiveness of intraoperative PINPOINT and Blue dye in identifying LNs defined as the proportion of LNs identified by PINPOINT and Blue dye respectively (confirmed as lymphoid tissue by histology) divided by the total number of LNs identified and excised.

#### **Secondary Variables**

LN detection rate with PINPOINT or Blue dye, defined as the proportion of cases in which at least one LN is identified with PINPOINT or Blue dye (confirmed as lymphoid tissue by histology).

Incidence of adverse events and adverse device events/effects of PINPOINT and Blue dye.

#### Other Variables

- Bilateral LN detection rate defined as the proportion of cases in which at least one LN is identified on right and left side of the pelvis.
- Proportion of LNs identified from following LCs.
- Anatomic distribution of LNs.

# Study Procedures and Assessments:

The following tests and procedures will be performed:

- · Vital signs, height, weight, demographics, surgical predictive factors.
- · Relevant medical history and underlying conditions.
- · Assessment of eligibility criteria.
- · Randomization to the B-P Arm or P-B Arm.
- · Imaging agent administration
- LN identification with PINPOINT and Blue dye followed by excision of all LNs.
- Documentation of LN mapping procedure.
- · Histological assessment of all excised lymph nodes
- · Concomitant medications
- · Assessment of surgical complications
- · Adverse events and adverse device effects
- Follow-up visits on date of discharge, and Day 30. Subjects with a discharge date later than Day 30 will have their last study visit on Day 30.



#### Sample Size and Statistical Analysis:

The FILM trial is a non-inferiority study comparing lymph node detection rates between Blue dye and PINPOINT. A sample size of approximately 150 evaluable subjects (to identify 525 LNs) is required to show the LN detection rate for PINPOINT is non-inferior to that with Blue dye with 80% power and a 5% 2-sided significance level with a 5% non-inferiority margin.

Both a modified Intent-to-Treat (mITT) and Per-Protocol (PP) analysis population will be utilized for the primary analysis. Analysis of the primary objective will be conducted using a 2-sided 95% confidence interval for the difference in proportions. A a non-inferiority test will be conducted using the PP and the mITT analysis populations. If and only if non-inferiority is claimed, a superiority test will be conducted using the mITT analysis population.<sup>3</sup> As a supporting analysis of the primary outcome, the analysis will also be repated using the as-treated (AT) population. The secondary objectives will be tested using a two -sided 5% significance level with a step-down multiplicity adjustment.

#### Study Duration:

The study is expected to begin in 2015 and complete enrollment in 18 months. Therefore, the study is expected to complete in 2017.



# **TABLE OF CONTENTS**

| PRO | TOCOL APPROVAL | 2 |
|---|---|---|
| PRO | TOCOL APPROVAL | 3 |
| PRO | TOCOL APPROVAL | 4 |
| PRO | TOCOL SUMMARY | 5 |
| ABB | REVIATIONS AND DEFINITIONS | 13 |
| 1 | INTRODUCTION AND BACKGROUND | 14 |
| 1.1.2<br>1.1.3 | Background Lymph Node Identification and Mapping. Endometrial and Cervical Cancer. Summary of Clinical Data for NIR Fluorescence Imaging with ICG for Lymphatic Mapping. Clinical Studies. | 14<br>14<br>15 |
| 1.2 | Potential Risks and Benefits to Human Subjects | 18 |
| 2 | STUDY OBJECTIVES | 19 |
| <b>2.1</b><br>2.1.1<br>2.1.2 | Objectives | 19 |
| 3 | INVESTIGATIONAL PLAN | 19 |
| 3.1 | Study Design Overview | 19 |
| 4 | SELECTION AND WITHDRAWAL OF SUBJECTS | 22 |
| 4.1 | Number of Subjects | 22 |
| 4.2 | Inclusion Criteria | 22 |
| 4.3 | Exclusion Criteria | 23 |
| 4.4 | Withdrawal of Subjects | 23 |
| 5 | RANDOMIZATION, BLINDING AND SUBJECT IDENTIFICATION PROCEDURES | 24 |
| <b>5.1</b><br>5.1.1 | RandomizationRandomization Procedure | |
| 5.2 | Subject Identification | 25 |
| 6 | STUDY TREATMENTS | 25 |
| 6.1 | Device Description | 25 |
| 6.2.1.<br>6.2.1.<br>6.2.1. | .2 Description of Investigational Product (IC2000) | 26<br>27<br>27 |
| 6.2.1 | .4 Labelling of IC2000 for Injection | 28 |



| 6.2.1. | | |
|---|---|---|
| - | Storage and administration of IC2000 for Injection | |
| 6.2.2. | | |
| 6.3 | Concomitant Treatment | 29 |
| 7 | RISKS/PRECAUTIONS | 30 |
| 7.1 | PINPOINT System – Endoscopes, Camera and Video Processor Illuminato | |
| | Unit | |
| 7.2 | Indocyanine Green (IC2000) | |
| 7.3 | Isosulfan Blue (Blue Dye) | |
| 8 | STUDY PROCEDURES | 32 |
| 8.1 | Schedule of Events | 32 |
| 8.2 | Baseline/Screening Procedures (Day -30 to Day 0) | 33 |
| 8.3 | Day 0 Procedures | |
| 8.3.1 <br>8.3.1.1 | Lymph Node Mapping Procedure | |
| 8.3.1. | | |
| 8.3.1. | | |
| 8.3.1.4 | Identification of Lymph Nodes with PINPOINT | 36 |
| 8.4 | Post-operative Follow-up Visits (Day of discharge to Day 30) | 38 |
| 8.5 | Histopathology of Excised LN | 38 |
| 9 | EVALUATION, RECORDING, AND REPORTING OF ADVERSE EVENTS | 39 |
| 9.1 | Definitions | |
| | Adverse Event (AE) | |
| | Adverse Device Effect (ADE)<br>Serious Adverse Event (SAE) | |
| | Unanticipated Adverse Device Effect (UADE) | |
| 9.2 | Adverse Event Descriptions | 40 |
| 9.2.1 | Intensity | 40 |
| | Relationship | 41 |
| 9.3 | Reporting and Evaluation of Serious Adverse Events and Unanticipated Adverse Device Effects | 41 |
| 9.4 | Follow-up for Adverse Device Effects and Adverse Events | 41 |
| 9.5 | Reporting of Technical Complaints/Device Deficiencies | 42 |
| 951 | Definitions | 42 |
| 9.5.2 | Reporting Procedures | 42 |
| 9.5.2<br><b>9.6</b> | Reporting Procedures ADEs Technical Complaints/Device Deficiencies that are UADEs | 42<br><b>42</b> |
| 9.5.2<br><b>9.6</b><br><b>10</b> | Reporting Procedures ADEs Technical Complaints/Device Deficiencies that are UADEs STATISTICAL CONSIDERATIONS | 42<br>42<br>43 |
| 9.5.2<br><b>9.6</b> | Reporting Procedures ADEs Technical Complaints/Device Deficiencies that are UADEs | 42<br>43<br>43 |



| 10.3 | Statistical Analysis | 43 |
|---|---|---|
| 10.4 | Sample Size Considerations | 44 |
| 10.5 | Data Sets to be Analyzed | |
| | Per-protocol (PP) | |
| | Modified Intent to treat (mITT) | |
| | As Treated (AT) | |
| 10.5. <del>-</del><br>10.6 | Secondary Objectives | |
| | Demographic and Baseline Data | |
| | Safety Variables and Analysis | |
| 10.7 | Handling of Missing Data | 48 |
| 10.8 | Pooling of Site Data | 48 |
| 11 | ESTIMATED DURATION OF THE STUDY | 48 |
| 12 | STUDY ETHICAL CONSIDERATIONS | 48 |
| 12.1 | Ethical Conduct of the Study | 48 |
| 12.2 | Informed Consent | 48 |
| 12.3 | Institutional Review Board, Ethics Committee, or Research Ethics Board (IRB) | 49 |
| 12.4 | Data and Safety Monitoring Board | 49 |
| 13 | ADMINISTRATIVE PROCEDURES | 49 |
| 13.1 | Sponsor's Responsibilities | |
| 13.1.1 | Public Disclosure of Clinical Trials | 49 |
| | Study Supplies | |
| | Investigator Training | |
| 13.1.3. | • | |
| 13.1.3. | J | |
| | Ongoing Communication of Safety Information During the Study | |
| | Records Retention | |
| 13.1.0<br>13.2 | Investigator's Responsibilities | |
| _ | Reporting and Recording of Study Data | |
| | Source Documentation | |
| | Study Devices and Imaging Agents | |
| | Records Retention | |
| 14 | DATA MANAGEMENT | 51 |
| 4 E | | |
| 15 | POLICY FOR PUBLICATION AND PRESENTATION OF DATA | 53 |



#### ABBREVIATIONS AND DEFINITIONS

ADE Adverse device effect

AE Adverse event AT As-treated

B-P BLUE-PINPOINT

CFR Code of Federal Regulations

CRF Case Report Form

CSF Color Segmented Fluorescence CT Computerized Tomography

DSMB Data and Safety Monitoring Board

EC Ethics Committee

FIGO International Federation of Gynecology and Obstetrics

FDA Food and Drug Administration

GCP Good Clinical Practice

GMP Good Manufacturing Practice

H&E Hematoxylin and eosin

HD High Definition

HAS Human serum albumin

IA Imaging agent

ICH International Conference on Harmonization

ICG Indocyanine Green

IRB Institutional Review Board IRC Image Review Committee

IV Intravenous

LC Lymphatic channel

LN Lymph node

MELD Model for end-stage liver disease

mITT Modified intent-to-treat

NCCN National Comprehensive Cancer Network

NDA New drug application

NIR Near-Infrared P-B PINPOINT-BLUE

PINPOINT PINPOINT Endoscopic Fluorescence Imaging System

PP Per-Protocol

REDCap Research Electronic Data Capture SADE Serious Adverse Device Effect

SAE Serious Adverse Event SLN Sentinel lymph node

US United States

UADE Unanticipated Adverse Device Effect

VIS Visible



#### 1 INTRODUCTION AND BACKGROUND

The study will be conducted in accordance with ethical principles that have their origin in the Declaration of Helsinki and in compliance with the protocol, Good Clinical Practice (GCP) and all applicable regulations.

# 1.1 Background

The purpose of this study is to assess the effectiveness of intraoperative PINPOINT Near Infrared Fluorescence Imaging in identification of lymph nodes (LN) in subjects with uterine and cervical malignancies who are undergoing lymph node mapping and to investigate the safety of interstitial injection of indocyanine green (IC2000) dye for intraoperative lymphatic mapping using PINPOINT Near Infrared Fluorescence Imaging.

## 1.1.1 Lymph Node Identification and Mapping

Identification of the tumor draining lymph nodes (LN has become an important step for staging cancers that spread through the lymphatic system. LN mapping involves the use of dyes and/or radiotracers to identify the LNs either for biopsy or resection and subsequent pathological assessment for metastasis. The goal of lymphadenectomy at the time of surgical staging is to identify and remove the LNs that are at high risk for local spread of the cancer

LN identification can be accomplished using several different methods, with the basic technique involving the injection of a tracer that identifies the lymphatic drainage pathway from the primary tumor<sup>6</sup>. The tracers used may be colored dyes (e.g. Isosulfan blue), or radioisotopes (e.g. technetium-99m) for intraoperative localization with a gamma probe; or, a combination of both. Recently, ICG using near-infrared (NIR) fluorescence imaging for visualization has emerged as a potentially effective method for several cancers including breast, skin (melanoma), cervical, endometrial, lung and gastrointestinal.

The PINPOINT system is an endoscopic NIR fluorescence imaging system used during minimally invasive surgical procedures. PINPOINT acquires NIR fluorescence images of an imaging agent (ICG) to allow for direct real time visual identification of a lymph node and/or the afferent lymphatic channel intraoperatively. ICG is a commonly used water soluble intravascular dye approved for human use in the United States and Canada. It has a peak spectral absorption at approximately 800 nm and can be used as a lymphatic NIR fluorophore. ICG binds primarily to globulins and to a lesser extent to lipoproteins and albumin<sup>§</sup>. In general, when injected interstitially, the protein binding properties of ICG cause it to be rapidly taken up by the lymph and moved through the conducting vessels to the LN<sup>§</sup>. The NIR fluorescent positive lymph nodes are represented on the PINPOINT screen in PINPOINT (green pseudo-color superimposed on white light image), SPY (black and white) or SPY CSF (color segmented fluorescence) mode.

#### 1.1.2 Endometrial and Cervical Cancer

Endometrial cancer is the most common gynecological cancer, and it is estimated that 52,630 new cases will be diagnosed in the United States (US)<sup>10</sup> and 6,000 new cases will be diagnosed in Canada in 2014<sup>11</sup>. Cervical cancer affects a lower number of women with 12,360<sup>12</sup> and 1,450<sup>11</sup> new cases estimated in the US and Canada respectively for 2014. The most important prognostic factor for subjects is accurate surgical staging, as lymph node status is a predictor of outcome and may influence treatment following surgery.



Identification of LNs and LN mapping for endometrial cancer is being evaluated as a method for surgical staging to be used in subjects with uterine confined tumors when there is no metastasis demonstrated by imaging studies and no obvious extrauterine disease 13. The current standard of care is to perform a complete or selective para-aortic lymphadenectomy for staging (FIGO) which can lead to morbidities such as lower extremity lymphedema and lymphocyst formation 4. Although the inclusion of pelvic and para-aortic lymphadenectomy in the surgical management is part of the FIGO staging, it remains controversial. Therefore, the decision about the extent of lymphadenectomy (e.g. pelvic nodes only or both pelvic and para-aortic nodes) done by the surgeon can still be based on the preoperative and intraoperative findings.

# 1.1.3 Summary of Clinical Data for NIR Fluorescence Imaging with ICG for Lymphatic Mapping

The imaging agent (IA), ICG (indocyanine green for injection, USP) 25 mg for Injection in the form of a sterile lyophilized powder containing indocyanine green with no more than 5% sodium iodide is approved by the FDA for determining cardiac output, hepatic function and liver blood flow, and for ophthalmic angiography via intravascular administration14,15. ICG is also approved under a 510(k) by the FDA for assessing blood flow and tissue perfusion in a variety of surgical and nonsurgical procedures16. ICG can be administered intravenously or intra-arterially. It absorbs light in the near-infrared region at 806 nm, and emits fluorescence (light) at a slightly longer wavelength, 830 nm. When injected intravenously, ICG rapidly and extensively binds to plasma proteins and is confined to the intravascular compartment with minimal leakage into the interstitium. This property makes ICG an ideal agent for the acquisition of high quality images of lymph nodes and lymphatic vessels (i.e., for NIR fluorescence lymphography).

#### 1.1.4 Clinical Studies

The Sponsor has not conducted any clinical trials on the use of intraoperative PINPOINT Near Infrared Fluorescence Imaging with ICG in identification and mapping of LN to date. However, 12 studies with performance and/or safety data using the Sponsor's fluorescence imaging devices or those with equivalent characteristics have been reported in the literature on the use of ICG in lymphatic mapping of gynecological cancers (<u>Table 1</u>).

**TABLE 1. Lymphatic Mapping Studies in Gynecological Cancers** 

| Author | Indication | Device | Summary |
|---|---|---|---|
| Furukawa et al., 2010 <sup>17</sup> | Cervical | PDE | ICG fluorescence imaging was used to identify SLN during sentinel node navigation surgery in cervical cancer patients. No allergic reactions to ICG were observed. |
| Crane et al., 2011 <sup>18</sup> | Cervical | Prototype<br>multispectral<br>fluorescence<br>camera system | Intraoperative lymphatic mapping and SLN detection was carried out in cervical cancer patients using ICG fluorescence imaging and patent blue dye. No side effects were noted after injection of ICG or patent blue dye. |
| Crane et al., 2011 <sup>19</sup> | Vulvar | Prototype<br>multispectral<br>fluorescence<br>camera system | Intraoperative transcutaneous lymphatic mapping was carried out in vulvar cancer patients in a comparison using ICG fluorescence imaging, 99m_Technetium-nanocolloid and patent blue dye. No side effects related to ICG injection were noted. |



| Author | Indication | Device | Summary |
|---|---|---|---|
| Holloway et al., 2012 <sup>20</sup> | Endometria<br>I | da Vinci Surgical<br>System | Retrospective comparison of results from lymphatic mapping of pelvic SLN using fluorescence NIR imaging of ICG and colorimetric imaging of Isosulfan blue dyes in women with endometrial cancer undergoing robotic-assisted lymphadenectomy. |
| Rossi et al 2012 <sup>21</sup> | Endometria<br>I | da Vinci Surgical<br>System | Sentinel lymph node (SLN) mapping with indocyanine green (ICG) detected by robotic near infrared (NIR) imaging is a feasible technique. |
| Schaafsma et al 2012 <sup>22</sup> | Cervical | Mini-FLARE | Eighteen consecutive early-stage cervical cancer patients scheduled to undergo pelvic lymphadenectomy were included. Prior to surgery, 1.6 mL of 500 μM ICG:HSA or 500 μM ICG alone was injected transvaginally in 4 quadrants around the tumor. The Mini-FLARE imaging system was used for intraoperative NIR fluorescence detection and quantitation. |
| Rossi et al<br>2013 <sup>23</sup> | Cervical or endometrial , Stage 1 | SPY Scope (7<br>subjects); da<br>Vinci (13<br>subjects) | Robotically assisted endoscopic NIR imaging after injection of ICG was used for LN mapping in patients with clinical stage 1 cervical or endometrial cancer. No AEs occurred. |
| Schaafsma et al 2013 <sup>24</sup> | Vulvar | Mini-FLARE | NIR fluorescence imaging for SLN biopsy was investigated and ICG vs ICG:HSA compared in a double-blind, randomized, non-inferiority trial of vulvar cancer patients. The study confirmed the feasibility of NIR fluorescence imaging for SLN mapping in vulvar cancer and found no advantage in using ICG:HSA over ICG alone. No AEs were associated with the use of ICG or ICG:HSA. |
| Jewell et al.,<br>2014 <sup>25</sup> | Endometria<br>I and<br>cervical | da Vinci Surgical<br>System | Robotically assisted endoscopic NIR imaging after injection of ICG was used for SLN mapping in patients with uterine and cervical malignancies |
| Sinno et al.<br>2014 <sup>26</sup> | Endometria<br>I or CAH | da Vinci Surgical<br>System | Comparison of NIR fluorometric imaging vs colorimetric imaging for SLN mapping in endometrial cancer |
| Plante et. al. 2015 <sup>27</sup> | Endometria<br>I and<br>cervical | PINPOINT<br>Endoscopic<br>System | Initial experience with PINPOINT Endoscopic NIR imaging for LN identification was reported. Study determined PINPOINT/ICG is an excellent and safe modality for SLN mapping with a very high (96%) detection rate. |
| How et. al. 2015 <sup>28</sup> | Endometria<br>I | da Vinci Surgical<br>System | Comparison of ICG, blue dye and 99mTc-SC mapping in patients undergoing robotic-assisted surgery. A mixture of all three modalities is feasible and provides good mapping. ICG was found to be superior to blue dye and comparable to 99mTc-SC and thus blue dye may not be essential for SLN detection. |

A total of 550 subjects with early stage gynecological cancers (cervical, endometrial and vulvar) have been reported in the literature as having undergone intraoperative SLN mapping with ICG fluorescence imaging. Table 2 lists the published studies including the number of subjects receiving ICG, the ICG dose, route of administration, SLN detection rate and safety results (when reported). All subjects receiving an injection of ICG are listed for studies that included co-administration of a colorimetric dye or radiotracer. Of the 12 studies, 7 specifically reported that there were no adverse reactions to the procedure. In 4 studies (Crane et al 2011; Furukawa et al 2010; Rossi et al, 2011, Plante et al. 2015), ICG fluorescence was used to identify SLNs in subjects with cervical or endometrial cancer <sup>17,19,21</sup> Detection rates ranged from 60% to 96%. In a study comparing ICG fluorescence and blue dye, Crane et al (2011) found that 89.7% of radioactively labelled SLNs in subjects with vulvar cancer could be detected by ICG fluorescence compared to 72.4% detected by blue dye<sup>18</sup>.

Schaafsma et al. compared the use of ICG and ICG conjugated to HSA for NIR fluorescence detection of SNs in subjects with early cervical cancer<sup>22</sup> and vulvar cancer<sup>24</sup>. In both studies, no difference in SLN detection rates was found between the ICG (6/9; 67% for cervical cancer and 9/12; 75% for vulvar cancer) and ICG: HSA groups (8/9; 89% for cervical cancer; 10/12; 83% for vulvar cancer) (p=0.13, cervical cancer; p=0.27, vulvar cancer).

Jewell et al. completed a retrospective, open label, single center study using NIR fluorescence imaging on the robotic platform with intracervical ICG injection for SLN detection in uterine and cervical malignancies<sup>25</sup>. A total of two hundred and twenty-seven cases were performed. When



ICG alone was used to map cases, 188/197 subjects mapped for a detection rate of 95% compared to 93% in cases in which both blue dye and ICG were used. Bilateral mapping was seen in 79% of ICG alone cases compared to 77% of cases using ICG and blue dye. The authors concluded that NIR fluorescence imaging on the robotic platform has a high bilateral detection rate and appears to be favorable to ICG dye alone, with blue dye combined with ICG unnecessary for SLN mapping.

How et al. recently completed a prospective study comparing NIR fluorescence using ICG, blue dye and technetium for SLN mapping in endometrial cancer<sup>28</sup>. A total of 100 subjects underwent SLN mapping with a mixture of ICG, blue dye and 99mTc-SC injected directly into the cervix. A total of 286 LNs were mapped (2.9 per subject). ICG had a significantly higher detection rate than blue dye both in unilateral (87% vs 71%) and bilateral (65% vs 43%) detection rates. The authors concluded that mapping with ICG is superior to blue dye and comparable to mapping with 99mTc-SC.

**TABLE 2 Lymphatic Mapping Studies in Gynecological Cancers** 

| Author | Type of<br>Cancer | Number<br>of<br>Patients | ICG<br>Concentration<br>(mg/ml) | Total Dose of ICG (mg) | Route of<br>Administration | Detection<br>Rate | Safety |
|---|---|---|---|---|---|---|---|
| Furukawa<br>et al., 2010 | Cervical | 10 | 5.00 | 1.0 | Cervical injection <sup>a</sup> | 83% | No allergic reactions |
| Crane et al., 2011 | Cervical<br>(1A1, 1B1,<br>IIA) | 10 | 0.50 | 0.50 Cervical injection | | 60% | No side effects reported |
| Crane et al., 2011 | Vulvar | 10 | 0.50 | 0.50 | Vulva<br>(peritumoral<br>injection) | 89.7% | No side effects related to intraoperative injection of ICG |
| Holloway et al., 2012 <sup>b</sup> | Endometria<br>I | 35 | 1.25 | 2.50 | Cervical injection <sup>a</sup> | 100% | Not reported |
| Rossi et al., | Cervical or | 3 | 0.50 | 0.50, 0.75 & | Cervical | 85% | No adverse |
| 2012 | endometrial<br>Stage 1 | al 17 | 0.50 | 1.5 injection <sup>d</sup> | | 88% | events reported |
| | ŭ | | | 1.00 | | | |
| Rossi et al.,<br>2012 | Endometria<br>I | 12 | 0.50 | 0.50 | Hysteroscopic endometrial | 33% | Not reported |
| | 17 0.50 1.00 Cervical Injection | | 82% | Not reported | | | |
| Schaafsma<br>et al., 2012 | Cervical<br>(1B1) | 9 | 0.38 | 0.62 | 0.62 Cervical <sup>a</sup> | | Not reported |
| Schaafsma<br>et al., 2013 | Vulvar | 12 | 0.38 | 0.62 | Vulva<br>(peritumorally or<br>around excision<br>scar) | 75% | No adverse reactions reported |
| Jewell et al.<br>2014 | Endometria<br>I and<br>cervical | 227 | 1.25 | 2.50 | Cervical<br>Injection | 100% | Not reported |
| Sinno et al.,<br>2014 | Endometria<br>I or CAH <sup>e</sup> | 38 | 1.25 | 5.00 | Cervical injection <sup>c</sup> | 78.9% | Not reported |
| Plante et al.<br>2015 | Cervical or<br>endometrial<br>Stage 1 | 50 | 1.25 | 5.00 | Cervical<br>Injection | 96% | No adverse events reported |



| Author | Type of<br>Cancer | Number<br>of<br>Patients | ICG<br>Concentration<br>(mg/ml) | Total Dose of<br>ICG (mg) | Route of<br>Administration | Detection<br>Rate | Safety |
|---|---|---|---|---|---|---|---|
| How et al.<br>2015 | Endometria<br>I | 100 | 0.25 | 0.1 | Cervical<br>Injection | 96% | No adverse events reported |

a Injection into 4 quadrants of the cervix (3, 6, 9 and 12 o'clock positions)

Based on the data available from clinical studies, this Phase III study has been designed to demonstrate the effectiveness of intraoperative PINPOINT Near Infrared Fluorescence Imaging in lymphatic mapping and to assess the safety of interstitial injection of ICG for intraoperative lymphatic mapping.

# 1.2 Potential Risks and Benefits to Human Subjects

Currently the PINPOINT system is classified by the United States Food and Drug Administration (FDA) as a Class II medical device with a Product Code of GCJ. PINPOINT for the purposes of fluorescence angiography is not identified as a significant risk device on the FDA Information Sheet titled "Significant Risk and Non-significant Risk Medical Device Studies". PINPOINT is a commercially available product in the United States (US) and Canada PINPOINT has a 510(k) clearance from the FDA and is licensed in Canada with the following indication:

"The PINPOINT system is intended to provide real-time endoscopic visible and near infrared fluorescence imaging. PINPOINT enables surgeons to perform routine visible light endoscopic procedures as well as further visually assess vessels, blood flow and related tissue perfusion with near infrared imaging during minimally invasive surgery".

Note: PINPOINT has not yet been classified by the FDA or Health Canada for the purposes of lymphatic mapping.

The imaging agent, ICG, is approved for human use by the FDA and Health Canada. In this study, investigational ICG (IC2000) will be administered interstitially for the visualization of LN and LC. The safety of interstitial administration of investigational IC2000 for NIR fluorescence imaging to identify LN has not been studied. However, safety data from published studies reported above combined with the well-established safety profile for ICG after intravenous or intra-arterial injection support an acceptable risk/benefit ratio for interstitial administration of ICG. The most serious risk of ICG when administered intravenously in humans, is anaphylactic death, which has been reported following ICG administration during cardiac catheterization.

These and other risks of the PINPOINT system in humans are described further in Section 7, Risks/Precautions. For additional information, please refer to the PINPOINT Operator's Manual<sup>16</sup>.

b Retrospective study

c Injection into cervix at 3 and 9 o'clock positions with 1 cc deep in the stroma and 1 cc submucosally on the right and left of cervix for a total volume of 4 ml

d Injection 1 cm into cervical stroma at 3 and 9 o'clock positions

e Complex Atypical Hyperplasia

f Intraoperative bilateral detection rate

# FILM

## 2 STUDY OBJECTIVES

## 2.1 Objectives

## 2.1.1 Primary Objectives

The primary objective of this study is to assess the effectiveness of intraoperative PINPOINT Near Infrared Fluorescence Imaging in identification of LNs in subjects with uterine and cervical malignancies who are undergoing LN mapping.

## 2.1.2 Secondary Objectives

- To evaluate the effectiveness of PINPOINT and Blue dye in the identification of at least one LN (confirmed to be lymphoid tissue) per subject.
- To evaluate the effectiveness of PINPOINT and Blue dye in the identification of bilateral LNs (confirmed to be lymphoid tissue).
- To assess the safety of interstitial injection of ICG for intraoperative lymphatic mapping.
- To determine the proportion of LNs identified from following LCs.
- To find the anatomic distribution of LNs.

# 3 INVESTIGATIONAL PLAN

# 3.1 Study Design Overview

This is a randomized prospective, open label, multicenter study to assess the safety and effectiveness of PINPOINT Near Infrared Fluorescence Imaging (PINPOINT) in identification of LN in subjects with uterine and cervical malignancies who are undergoing LN mapping. This is a non-inferiority within-subject comparison study to determine the effectiveness of PINPOINT in the identification of LNs compared to LNs identified with Blue dye. Approximately 150 subjects will be enrolled at up to 10 centers in North America. Prior to enrolling study subjects, participating surgeons at each center will be trained to perform intraoperative identification and mapping of LNs with ICG and Blue dye. Participating surgeons will be required to have completed at least 10 LN mapping procedures with a minimum of 3 LN mapping cases performed with PINPOINT prior to the initiation of enrollment.

## Screening:

Subjects diagnosed with International Federation of Gynecology and Obstetrics (FIGO) clinical stage I endometrial or cervical cancer scheduled for surgery that includes clinically indicated LN mapping will be evaluated at baseline to determine if they meet the inclusion/exclusion criteria of the protocol. Subjects will be assessed to determine overall health status including demographics, vital signs, diagnosis and relevant medical history/underlying conditions. Eligible subjects who provide informed consent will be considered for inclusion into the study.



**FIGURE 1. Group Assignment and Randomization** 



Day 0:

On the day of surgery, subjects will be randomized (1:1) to either the BLUE-PINPOINT (B-P) Arm or the PINPOINT-BLUE (P-B) Arm. Subjects in each arm will be randomized according to an independently generated randomization scheme to undergo lymphatic mapping with Blue dye first followed by mapping with PINPOINT (B-P Arm) or to undergo lymphatic mapping with PINPOINT first followed by mapping with Blue dye (P-B Arm).

PINPOINT® for Lymph Node Mapping Clinical Study Protocol PP LNM 01



Eligible subjects who have provided informed consent will be enrolled in the study upon randomization on the day of surgery (Day 0). Minimally invasive surgery will be performed according to the surgeon's standard practice.

The cervix will be injected four (4) times with a 1 ml solution of Blue Dye (1% Isosulfan blue; 10 mg/ml) for a total dose of 40 mg Blue Dye) and four (4) times with 1 ml of a 1.25 mg/ml solution of IC2000 for a total dose of 5 mg IC2000. The injection of Blue dye and IC2000 will occur while the subject is under anesthesia in the operating room.

In order to minimize the spillage of blue dye or ICG interfering with the mapping procedure when LNs are excised, mapping will be performed on one side of the pelvis followed by the other side and mapping with both Blue dye and PINPOINT will be performed prior to the excision of any LNs.

Subjects randomized into the B-P Arm will be administered Blue dye first followed by the administration of IC2000 and undergo LN mapping with Blue dye first followed by mapping with PINPOINT. LN mapping with Blue dye will be performed until the investigator identifies all blue nodes or determines that blue nodes cannot be identified. Once complete, the Investigator will begin mapping with PINPOINT until all 'IC2000' nodes are identified or the investigator determines that 'ICG' nodes cannot be identified. Once mapping with both Blue dye and PINPOINT have been completed and documented, all LNs identified with Blue dye or PINPOINT will be excised.

Subjects randomized into the P-B Arm will be administered IC2000 first followed by the administration of Blue dye and undergo LN mapping with PINPOINT first followed by mapping with Blue dye. LN mapping with PINPOINT will be performed until the investigator identifies all 'IC2000' nodes or determines that 'IC2000' nodes cannot be identified. Once complete, the Investigator will begin mapping with Blue dye until all 'blue' nodes are identified or the investigator determines that 'blue' nodes cannot be identified. Once mapping with both PINPOINT and Blue dye have been completed and documented, all LNs identified with PINPOINT or Blue dye will be excised.

LN mapping for Clinical Stage I endometrial cancer will be performed according to the NCCN Guidelines for Uterine Neoplasms, LN Algorithm for Surgical Staging of Endometrial Cancer; and LN mapping for Clinical Stage I cervical cancer will be performed according to the NCCN Guidelines for Cervical Neoplasms, Surgical/LN Mapping Algorithm for Early-Stage Cervical Cancer 1.2.

The surgeon will identify LN based on direct visualization with white light for blue dye or PINPOINT for IC2000.

# LN Mapping with PINPOINT:

Intraoperative identification of LNs with IC2000 will be based on the following criteria:

- Direct visual identification of a node by NIR fluorescence with IC2000 using PINPOINT.
- Visibly or palpably abnormal LNs designated as palpable masses and excised regardless of visible fluorescence.

.

Mapping will be considered complete when all nodes meeting any of the criteria above are identified and documented and the surgeon has scanned the full 360-degree area within the abdominal cavity. Fluorescent ducts should be followed in both directions in order to identify LNs to be excised.

PINPOINT® for Lymph Node Mapping Clinical Study Protocol PP LNM 01



LN Mapping with Blue dye:

Intraoperative identification of LNs with Blue dye will be based on the following criteria:

- Direct visual identification of a node stained with Blue dye.
- Visibly or palpably abnormal LNs designated as palpable masses and excised regardless
  of visible blue dye.

Mapping will be considered complete when all nodes and channels meeting any of the criteria above are identified and documented and the surgeon has scanned the full 360-degree area within the abdominal cavity. Blue ducts should be followed in both directions in order to identify LNs to be excised.

#### Classification of LNs:

All LNs identified will be classified as:

- 1. Fluorescent only
- 2. Blue only
- 3. Both (Fluorescent and blue)
- 4. Abnormal or palpably hard
- 5. Non-stained node found at origin or termination of fluorescent duct
- 6. Non-stained node found at origin or termination of blue duct
- 7. Non-stained node found at origin or termination of fluorescent and blue duct

Effectiveness of intraoperative Blue dye in identifying of LN will be based on the proportion of LNs identified by visualization of blue dye under white light and confirmed as lymphoid tissue by histology divided by the total number of LNs identified and excised.

Effectiveness of intraoperative PINPOINT in identifying of LN will be based on the proportion of LNs identified by PINPOINT and confirmed as lymphoid tissue by histology divided by the total number of LNs identified and excised.

Details of the surgery, including intraoperative findings will be documented. Surgical data will be collected including the ability to identify LNs, the number of LNs identified and removed, the ability to unilaterally and bilaterally map LNs, and the anatomical location and distribution of identified LNs. Failed mapping is defined as no LNs detected.

## Follow-up and Post-operative Complications:

All Subjects will have standard of care assessments throughout the study according to the hospital/institution's standard procedures as well as study specific visits to monitor occurrence of any adverse events/adverse device effects on the date of discharge and Day 30 (±7 days). All subjects will be followed to monitor occurrence of adverse events up to Day 30 (±7 days) post-surgery. All adverse events will be followed up to Day 30 (±7 days). Adverse events thought to be related to the use of PINPOINT or to the LN mapping procedure will be followed until resolution or deemed chronic.

#### 4 SELECTION AND WITHDRAWAL OF SUBJECTS

## 4.1 Number of Subjects

Approximately 150 subjects will be enrolled in the study (See Section 10.4).

#### 4.2 Inclusion Criteria



To be eligible for the study, a subject must fulfill all of the following criteria:

- 1. Be 18 years of age or older
- 2. Have either of the following diagnoses and surgical plan:
  - a. FIGO Clinical stage I endometrial cancer undergoing minimally invasive hysterectomy with lymphatic mapping
  - b. FIGO Clinical stage IA cervical cancer ≤ 2 cm undergoing minimally invasive hysterectomy, trachelectomy or conization with lymphatic mapping. Note: Subjects with clinical Stage IA1 cervical cancer without lympho vascular space involvement (LVSI) and negative margins on cone biopsy are not to be included.
- 3. Negative nodal status (N0)
- 4. Subjects with negative metastatic involvement (M0)
- 5. Subjects of child-bearing potential must not be pregnant or lactating and must have a negative pregnancy test at Day 0
- 6. Have signed an approved informed consent form for the study
- 7. Be willing to comply with the protocol

#### 4.3 Exclusion Criteria

A subject meeting any of the following criteria will be excluded from the study:

- 1. Have had prior dissection and/or radiation in pelvis
- 2. Advanced cervical or endometrial cancer, T3/T4 lesions
- 3. Diagnosis of cervical cancer with a tumor size greater than 2 cm
- 4. Locally advanced cervical or uterine cancer
- 5. Metastatic cervical or uterine cancer
- 6. Known allergy or history of adverse reaction to ICG, iodine or iodine dyes
- 7. Known allergy or history of adverse reaction to Blue dye (Isosulfan blue) or triphenylmethane
- 8. Hepatic dysfunction defined as MELD Score > 12
- 9. Renal dysfunction defined as serum creatinine ≥ 2.0 mg/dl
- 10. Subjects who have participated in another investigational study within 30 days prior to surgery
- 11. Pregnant or lactating subjects
- 12. Subjects who, in the Investigator's opinion, have any medical condition that makes the subject a poor candidate for the investigational procedure, or interferes with the interpretation of study results

## 4.4 Withdrawal of Subjects

Subjects can voluntarily withdraw (or be withdrawn) at any time during the study. Investigators may withdraw a subject from the study because:



- A new health condition, diagnosis or finding appears that is suspected to require care or medication prohibited by the protocol.
  - o e.g., the planned surgical procedure is modified to a procedure prohibited by the protocol.
- The subject has unacceptable adverse events.
- It is in the subject's best interest according to the Investigator's clinical judgment.

If a subject is prematurely withdrawn from the study, the reason(s) for withdrawal must be recorded on the relevant page of the subject's Study Completion case report form (CRF).

Subjects who discontinue the study prematurely will not be replaced.

The Sponsor may stop the study at any time.

## 5 RANDOMIZATION, BLINDING AND SUBJECT IDENTIFICATION PROCEDURES

#### 5.1 Randomization

Subjects will be prospectively randomized into the FILM Clinical Trial. Randomization will occur on the day of surgery. Prior to surgery, the subject will have provided written informed consent, completed all baseline procedures and met the requirements of inclusion and exclusion criteria. Randomization should be performed as closely as possible to the mapping procedure to minimize the incidence of dropout.

Subjects will be randomly assigned on a one to one (1:1) basis to either the B-P Arm (LN mapping with Blue dye followed by LN mapping with PINPOINT) or the P-B Arm (LN mapping with PINPOINT followed by LN mapping with Blue dye). Randomization will be stratified by study site. Permuted block randomization will be performed within strata. To minimize the opportunity for the sequence to be predicted, the block size will be variable and randomly chosen from small multiples of 2 (i.e. 2, 4 or 6). The randomization schedules will be generated in advance using a computerized random number generator. Investigational sites will not have access to the randomization schedules.

Randomization will be accomplished using a secure web-based software (REDCap) supported by the Data Coordinating Center. Treatment assignment is made only after verification of proper informed consent execution and study eligibility.

## 5.1.1 Randomization Procedure

The study coordinator or a designee will verify that the subject is eligible and that informed consent has been obtained prior to initiating the randomization process. On the day of surgery the study coordinator will log onto the REDCap system and, after confirming the subject's



eligibility, will enroll a subject and obtain the randomization assignment. The study coordinator will then disclose the randomization assignment to the Investigator. As this is a within-subject comparison study, the investigator cannot be blinded to the use of Blue dye or PINPOINT device. All subjects will be blinded to their randomization assignment until after the procedure.

A subject is not randomized until randomization has been assigned by REDCap. The randomization procedure should not be initiated unless the study coordinator confirms that a subject is eligible and verifies baseline information. If any deviations occur (errors such as assigning incorrect randomization), the clinical site will be required to contact the Sponsor and await guidance on how to proceed.

If, at any time after randomization, the subject becomes ineligible or withdraws, the subject is still considered randomized. If an intraoperative decision is made to perform a procedure other than what was intended, the subject will be categorized with respect to the definitions outlined for the analysis populations (see the Statistical Methods Section 10.5).

# 5.2 Subject Identification

Screening ID Number: All subjects screened for the study shall be assigned a 5-digit "screening" number on the Screening Log and if they are randomized, will subsequently be assigned a Subject Enrollment Number in the electronic data capture system. The Screening Identification Number shall be unique and categorize a subject in sequence of screening by an "S" followed by a 5-digit number. The first 2 digits identify the site and the last three digits identify the subject. For example, the first subject screened at site 01 is identified as screening number S- 01001. The screening log shall be maintained by the site to identify those subjects that have failed screening with the reason why they did not qualify for enrollment. The screening number will be assigned sequentially within each study center in order of subject presentation for screening.

Enrolled Subject ID Number: Once a subject is randomized, they will be assigned a Subject Enrollment Number which is also a 5-digit number. The first two digits of the Subject Enrollment Number identify the site and the last three digits identify the subject. Each site will be given a Site Identification Number. For example, the first subject randomized at site 03 is identified as subject 03-001, the next subject as 03-002, etc.

Subjects who sign an informed consent form but are not randomized are considered screen failures. These subjects must be entered on the Screening Log but do not receive a subject number. The reason for non-enrollment must be documented on the log.

#### **6 STUDY TREATMENTS**

## **6.1 Device Description**

PINPOINT is an endoscopic fluorescence imaging system for high definition (HD) visible (VIS) light and near-infrared (NIR) fluorescence imaging. PINPOINT includes the following components:

- A surgical endoscope optimized for VIS/NIR illumination and imaging, which is available in different diameters, lengths and directions of view (Model: SC9104, SC9134).
- A camera head that is also optimized for VIS/NIR imaging and mounts to the endoscope eyepiece (Model: PC9002).
- A flexible light guide cable (Model: PC9004).

# PINPOINT® for Lymph Node Mapping Clinical Study Protocol PP LNM 01



 An endoscopic Video Processor / Illuminator (VPI) capable of providing VIS/NIR illumination to the surgical endoscope via a flexible light guide cable, and the image processing required to generate simultaneous, real-time HD video color and NIR fluorescence images (Model: PC9001).

PINPOINT is designed to be connected to a medical-grade HD color monitor, such as those normally used in surgical endoscopy.

PINPOINT is connected to a high-definition medical video recorder (Sony HVO-1000) that allows the capture of still images and video during operation.

PINPOINT acquires NIR fluorescence images of an imaging agent (IC2000) to allow for visual assessment of vessels, blood flow and related tissue perfusion during minimally invasive surgery. For the purpose of this study, PINPOINT will be used for visual identification of LNs during LN mapping procedures.

The PINPOINT Operator's Manual <sup>16</sup> describes the contents, use and storage of the PINPOINT PAQ's. Instructions for preparation, handling and administration of Investigational ICG (IC 2000) are provided in <u>Section 8.3.1.2</u>.

PINPOINT allows simultaneous display of multiple images. Real time NIR fluorescence video images are acquired by using the imaging agent and may be viewed in two ways:

PINPOINT image: NIR fluorescence is superimposed in pseudo-color (green) on a white light

image

SPY image: A black and white NIR fluorescence image is displayed

CSF: A high-definition, white light image is displayed in

gravscale with NIR fluorescence overlaid on a color scale. Increasing

fluorescence levels transition from blue through yellow to red.

PINPOINT also operates as a conventional endoscopic imaging system and provides illumination for real-time color (white light) HD video imaging in the area of interest.

PINPOINT is a commercially available product in the United States (US) and Canada. PINPOINT has a 510(k) clearance from the FDA and a Health Canada license with the following indication:

"The PINPOINT system is intended to provide real-time endoscopic visible and near infrared fluorescence imaging. PINPOINT enables surgeons to perform routine visible light endoscopic procedures as well as further visually assess vessels, blood flow and related tissue perfusion with near infrared imaging during minimally invasive surgery".

PINPOINT is manufactured by Novadaq Technologies Inc. (Novadaq). Please refer to the current version of the PINPOINT Operator's Manual<sup>16</sup> for a full description and specifications of the system.

In this study, the use of PINPOINT for visual identification of lymph nodes via interstitial injection of ICG is investigational.

#### **6.2 Imaging Agent Description**

## 6.2.1 Indocyanine Green IC2000



# 6.2.1.1 Overview and Pharmacokinetics of Investigational Product

ICG was originally approved by the FDA for human medical use in 1959 for use in determining cardiac output, hepatic function and liver blood flow. In 1975, a NDA Supplement was approved for ICG for use in ophthalmic angiography. In 2005, ICG was approved under a 510K for assessing blood flow and tissue perfusion in a variety of surgical and non-surgical procedures. Over the past 50 years ICG has been marketed in the United States and has demonstrated an excellent safety profile. ICG has received approval from Health Canada (DIN 02014793) in 1994 for human medical use as a diagnostic agent, and is classified as an "Ethical" drug.

ICG absorbs light in the near-infrared (NIR) region at 806 nm and emits fluorescence (light) at a slightly longer wavelength, 830 nm. After injection, ICG rapidly binds to blood proteins primarily lipoproteins and to a lesser extent globulins and albumin and drains into the lymphatic system without extravasation enabling sensitive non-invasive visualization of LN and lymphatic architecture. Within minutes after intravenous injection, ICG is cleared by the liver and excreted into the bile<sup>24</sup>. Since lymph fluid flows into the venous blood stream through the subclavien veins<sup>9</sup>, it is assumed that, after interstitial injection, ICG drains with lymph fluid into the circulatory system where it is then cleared by the liver and excreted in the bile. Although formal pharmacokinetic studies have not been performed with non-intravenous routes of administration, after intradermal injection in mice, ICG was shown to be taken up by lymphatic vessels and cleared within 48 hours<sup>29,30</sup>. Another study using ICG conjugated to human serum albumin (HSA) in rabbits found ICG is efficiently taken up by the lymphatic vessels and cleared within 24 hours after peritumoral injection<sup>31</sup>. Chi et al. investigated the use of ICG for LN mapping in 5 mice, 10 rabbits and 22 breast cancer subjects and found LNs are identifiable 3-5 minutes after injection with the occurrence of peak fluorescence intensities varying with the dose of ICG and occurs between 10 and 90 minutes<sup>32</sup>.

# 6.2.1.2 Description of Investigational Product (IC2000)

The chemical name of the investigational drug, indocyanine green is 1 *H*-Benz[e]indolium, 2-[7-[1,3-dihydro-1,1-dimethyl-3-(4-sulfobutyl)-2*H*-benz[e]indol-2-ylidene]-1,3,5-heptatrienyl]-1,1-dimethyl-3-(4-sulfobutyl)-,hydroxide, inner salt, sodium salt. ICG has a molecular weight of 774.96 daltons and will be administered with an interstitial injection into the cervix.

The imaging agent, IC2000 (indocyanine green, USP) is provided in the form of a sterile lyophilized powder containing 25 mg ICG with no more than 5% sodium iodide. IC2000 is packaged with aqueous solvent consisting of sterile Water for Injection, which is used to reconstitute the ICG. When injected, ICG rapidly and extensively binds to plasma proteins (primarily lipoproteins and globulins) with minimal leakage through vessel walls. This property makes ICG an ideal agent for the acquisition of high quality images of LNs and s (i.e., for NIR fluorescence lymphography). Note: The use of IC2000 in this study is investigational.

#### 6.2.1.3 Chemistry and Manufacturing

Investigational IC2000 is supplied as a 25 mg sterile lyophilized green powder in a glass vial with a grey stopper and grey over seal. The product is stored at 20°C to 25°C (68° to 77° F). IC2000 is manufactured by Patheon (Patheon Italia S.p.A., 2° Trav. SX Via Morolense, 503013 Ferentino- Italy) and, like commercially available ICG, IC2000 is tested according to the USP monograph for Indocyanine green for Injection.

PINPOINT® for Lymph Node Mapping Clinical Study Protocol PP LNM 01



IC2000 was manufactured in full compliance with the FDA's current Good Manufacturing Practice (cGMP) for Finished Pharmaceuticals-standards at 21 CFR Part 211 and meets all GMP requirements for Health Canada.

## 6.2.1.4 Labelling of IC2000 for Injection

IC2000 is labeled according to US and Canadian regulatory requirements with the following information:

- IC2000 (indocyanine green for injection, USP), 25 mg lyophilized ICG
- Sterile
- Protocol No.: PP LMN 01
- Directions for use: Refer to Clinical Protocol
- Store at: 20–25°C (68-77°F)
- Lot: 14GRF03
- EXP.: May 2016
- CAUTION—New drug Limited by Federal (or United States) law to investigational use.
- Investigational drug to be used only by a qualified investigator.
- Sponsor: Novadaq Technologies Inc. 13155 Delf Place, Unit 250, Richmond, BC, Canada, V6V 2A2 1.844 6682327

## 6.2.1.5 Packaging and Distribution of IC2000

IC2000 will be packaged into investigational PINPOINT LN Mapping Kits as described below and distributed by the study Sponsor (Novadaq). Each LN-mapping procedure kit is indicated for use exclusively with PINPOINT and should only be used for the purposes of this study.

Each PINPOINT LN Mapping kit contains:

- One single use 25 mg vial of sterile IC2000, USP
- Two single use 10 ml ampules of sterile Aqueous solvent
- Four 3 ml syringes, sterile
- Two 10 ml syringes, sterile
- Two Lure-lock 10 ml syringes with controlled handle
- Four Spinal needles, 22G, 3.5 inch, sterile
- Labels for syringes

All information included on the investigational IC2000 for Injection vial labels will appear on the kit labels along with a description of the contents of the kit. Each kit will bear a unique serial number and will meet regulatory requirements necessary for each participating country.

# 6.2.1.6 Storage and administration of IC2000 for Injection

IC2000 will be stored at 20°C to 25°C (68° to 77° F) in a secure locked area, accessible to authorized personnel only. IC2000 will be stored, handled, prepared and administered by qualified, trained personnel only as described in <a href="Section 8.3.1.2">Section 8.3.1.2</a>.



## 6.2.2 Blue Dye (Isosulfan Blue)

The Blue dye (Isosulfan Blue Injection, 1% aqueous solution) a sterile and pyrogen-free 5 ml single-use vial<sup>33</sup>. Isosulfan blue is supplied as a 1% aqueous solution in a phosphate buffer and is approved under an ANDA by the US FDA for the identification of lymphatic vessels draining the region of injection, lymphography, and identification of lymph node involvement by primary and secondary neoplasms. Isosulfan blue will be obtained from commercially available sources and is approved for subcutaneous injection.

#### 6.2.2.1 Storage and administration

Blue dye will be stored at 20°C to 25°C (68° to 77° F) in a secure locked area, accessible to authorized personnel only. Blue dye will be stored, handled, prepared and administered by qualified, trained personnel only as described in Section 8.3.1.1.

# Installation, Training and Storage

PINPOINT will be installed by Novadaq representatives. The Investigator(s) and study staff shall be required to participate in training on the operational and procedural use of PINPOINT as it relates to the conduct of this study. Training will be provided by Novadaq.

Prior to enrollment, participating Investigator surgeons must be experienced with LN mapping procedures (i.e. performed a minimum of 10 LN mapping procedures) with a minimum of 3 LN mapping cases performed with PINPOINT prior to initiation of enrollment.

Investigator surgeons new to this technique will receive training consisting of the following:

- Didactic training on product and procedure.
- Hands on training session with clinical specialists on site.
- Guidance on use of the system and interpretation of the images with a clinical educator during a minimum of 10 cases prior to study enrollment.

Supporting personnel operating and cleaning PINPOINT will also receive training and be familiar with all applicable aspects of the operation and cleaning of the system.

PINPOINT shall be stored at room temperature in a secure and limited access area available to study staff.

#### 6.3 Concomitant Treatment

Any concomitant medications the subject is receiving at the start of the study (Day 0) or given for any reason during the study must be recorded in the CRF and source documents with the



exception of routine medications given for preparation of surgery, during surgery and postoperative care. These include but are not limited to the following:

- Sedatives and anesthetics
- Anticoagulants
- Prophylactic antibiotics
- Anti-emetics
- Routine post-operative pain medications

The drug name, start and stop dates, indication, dose, frequency and route information will be recorded for concomitant medications.

Other surgical and diagnostic procedures concomitant to the laparoscopic hysterectomy, trachelectomy, conization and lymphatic mapping procedure that take place during the study must be recorded in the CRF and in the source document, including start and stop dates.

# 7 RISKS/PRECAUTIONS

Refer to the PINPOINT Operator's Manual for a full description of the risks and precautions associated with all components of PINPOINT. The entire PINPOINT Operator's Manual should be read before using PINPOINT<sup>16</sup>. Failure to follow the instructions and warnings in the manual may result in unsafe operation of the system and/or injury to the subject or operator.

Refer to the Isosulfan Blue prescribing information for a full description of risks and precautions associated with the use of Isosulfan Blue<sup>33</sup>. The entire package insert should be read before using Isosulfan blue. Failure to follow instructions and warnings may result in injury to the subject.

## 7.1 PINPOINT System - Endoscopes, Camera and Video Processor Illuminator Unit

Currently, PINPOINT is classified by the FDA as a Class II medical device with a Product Code of GCJ. PINPOINT for the purposes of fluorescence angiography is not identified as a significant risk device on the FDA Information Sheet titled "Significant Risk and Non-significant Risk Medical Device Studies".

The use of PINPOINT for LN mapping is investigational. PINPOINT should only be used in accordance to its approved Indication for Use or in accordance to the study procedures described in this protocol.

# 7.2 Indocyanine Green (IC2000)

IC2000 will be injected directly into the cervical submucosa and stroma; and will not be administered intravenously. Additionally, the subject is anesthetized and the cervix and uterus are removed as part of the surgical procedure. Therefore the risks associated with injection into the cervix are expected to be lower than those associated with intravenous administration. Based on the clinical information for systemic ICG administration, the risks and precautions are discussed below.

PINPOINT® for Lymph Node Mapping Clinical Study Protocol PP LNM 01



Severe allergic reaction (affects fewer than one in every 10,000 subjects) with symptoms that could include the following: tightness in the throat, itchy skin, blotchy skin, rash, coronary artery spasm, facial edema, breathing difficulties, tightness and/or pain in the chest, faster heartbeat, a fall in blood pressure and shortness of breath, cardiac arrest, restlessness, nausea, feeling of warmth, flushes, hypereosinophilia<sup>15</sup>.

The possibility of an allergic reaction is greater in subjects with extremely serious kidney failure. To minimize the risk of an allergic reaction, all subjects with renal dysfunction are excluded as well as subjects with a known allergy to iodine, ICG or iodine dyes 15.

IC2000 contains sodium iodide and should be used with caution in subjects who have a history of allergy to iodides or iodinated imaging agents. Anaphylactic or urticarial reactions have been reported in subjects with and without history of allergy to iodides. Anaphylactic deaths have been reported following ICG administration during cardiac catheterization<sup>14</sup>.

Radioactive iodine uptake studies should not be performed for at least 1 week following IC2000 administration 14,15.

Animal reproduction studies have not been conducted with ICG or IC2000. It is not known whether ICG or IC2000 can cause fetal harm when administered to a pregnant woman or can affect reproduction capacity. It is not known whether ICG or IC 2000 is secreted in human milk. Women who are pregnant or lactating are excluded from this study.

# 7.3 Isosulfan Blue (Blue Dye)

Similar to the administration of IC2000 in this study, Isosulfan blue will be directly injected into the cervical submucosa and stroma. The subject will be anaesthetized and the cervix and uterus are removed as part of the surgical procedure.

Severe anaphylactic reactions have occurred after injection of Isosulfan blue (approximately 2% of subjects). Manifestations include respiratory distress, shock, angioedema, urticarial and pruritus. Reactions are more likely to occur in subjects with a history of bronchial asthma, or subjects with allergies or drug reactions to triphenylmethane dyes.

Isosulfan blue interferes with measurements of oxygen saturation by pulse oximetry and methemoglobin by gas analyzer.

The use of Isosulfan blue may result in transient of long-term (tattooing) blue coloration.

It is not known whether Isosulfan blue can cause fetal harm when administered to a pregnant woman or can affect reproduction capacity. It is not known whether Isosulfan blue is secreted in human milk. Women who are pregnant or lactating are excluded from this study.



# **8 STUDY PROCEDURES**

## 8.1 Schedule of Events

**Table 3** Schedule of Events

| | Baseline | Day 0 (Operative Phase) | | | | |
|---|---|---|---|---|---|---|
| Procedure | (Day -30 to Day<br>0) | Pre-OP | Intra-Op | Post-Op | Date of Discharge | Day 30 Phone call ( <u>+</u> 7 days) <sup>a</sup> |
| Informed consent | X | | | | | |
| Demography, Surgical risk factors | Х | | | | | |
| Vital signs, blood pressure, heart rate, height, weight | Х | | | | | |
| Pre-operative diagnosis | Х | | | | | |
| Pregnancy test | Х | | | | | |
| Inclusion/exclusion criteria | Х | | | | | |
| Serum sodium, bilirubin, creatinine and INR for MELD Score | Х | | | | | |
| Hemoglobin | Xq | | Xp | | | |
| Randomization | | Х | | | | |
| LN mapping with Blue dye | | | Х | | | |
| LN mapping with PINPOINT | | | Х | | | |
| Surgical Procedure | | | Х | | | |
| Documentation of LN mapping and surgical procedure | | | Х | Х | | |
| Concomitant medications and procedures | Х | Х | Х | Х | X | Х |
| Adverse events/adverse device effects | | Х | Х | Х | Х | Xc |
| Histopathological evaluation of Lymph<br>Nodes | | | Х | Х | | |

Subjects with a discharge date later than Day 30, will have the last study visit on Day 30.

Hemoglobin measurement at the time of mapping if the subject had any hypotensive events or blood loss over 500 ml at the time of mapping.

All subjects with adverse events thought to be related to the LN mapping procedure or the PINPOINT system will be followed until resolution or deemed chronic. Hemoglobin measurement must occur within 14 days prior to the day of surgery (Day -14 to day 0)



# 8.2 Baseline/Screening Procedures (Day -30 to Day 0)

After signing the informed consent form, subjects will be assigned a screening number (see Section 5.2) and be evaluated for eligibility into the study.

The following procedures will be conducted during the baseline assessment:

- Collection of demographics, surgical risk factors, pre-operative diagnosis
- Vital signs (heart rate and blood pressure), height and weight
- Serum tests (sodium, bilirubin, creatinine and INR) for MELD Score
  - The following calculator from the OPTN website should be used to calculate the MELD Score:

https://optn.transplant.hrsa.gov/resources/allocation-calculators/meld-calculator/

- Pregnancy test (urine test or institution standard of care) for subjects of childbearing potential on Day 0
- Hemoglobin measurement within 14 days prior to the date of surgery.

## 8.3 Day 0 Procedures

On the day of surgery, subjects will be randomized as described in <u>Section 5.1</u>. Subjects are considered enrolled upon randomization.

According to the randomization assignment, subjects randomized into the B-P Arm will be administered Blue dye first followed by the administration of IC2000. Subjects in the B-P arm will undergo LN mapping with Blue dye first followed by mapping with PINPOINT.

Subjects randomized into the P-B Arm will be administered IC2000 first followed by the administration of Blue dye and undergo LN mapping with PINPOINT first followed by mapping with Blue dye.

All subjects will undergo the appropriate surgical procedure (minimally invasive hysterectomy, trachelectomy or conization) according to the surgeon's standard practice. The surgical procedures include the following:

- Hysterectomy, Radical Hysterectomy
- Radical Trachelectomy
- Bilateral Salpingo-ophorectomy, Unilateral Salpingo-ophorectomy
- Ovarian Transposition
- Sentinel Lymph Node Mapping



- Pelvic Lymph Node Sampling
- Pelvic Lymph Node Dissection
- Para-aortic Lymph Node Sampling
- Para-aortic Lymph Node Dissection

All subjects will receive the hospital/institution and surgeon's standard pre-operative and post- operative care with the addition of any study specific requirements.

An intra-operative measurement of hemoglobin should be performed at the time of mapping if the subject experiences a hypotensive event requiring intraoperative management (e.g. use of vasopressors) or blood loss greater than 500 ml at the time of mapping.

Either during or immediately post-operatively, the details of the LN mapping procedure and surgical procedure will be documented. LN mapping data will be collected including the ability to identify LN, the ability to unilaterally and bilaterally map LN, and anatomical location and distribution of identified LN. Failed mapping is defined as no LN detected.

The following elements must be included and recorded in the case report form (CRF):

- Surgical time and estimated blood loss
- Dose of Blue dye administered
- Dose of IC2000 administered
- Details on injection technique
- Total number of LNs identified with PINPOINT
- Total number of LNs identified with Blue dye
- Total number of abnormal LNs identified (suspicious nodes)
- Total number of LNs excised
- Classification of LNs identified
- LNs anatomical location and distribution
- Pathological status of LNs excised
- Concomitant medications and procedures as described in Section 6.3
- Adverse events according to <u>Section 9</u>

# 8.3.1 Lymph Node Mapping Procedure

LN mapping for FIGO Clinical Stage I endometrial cancer will be performed according to the NCCN Guidelines for Uterine Neoplasms, SLN Algorithm for Surgical Staging of Endometrial Cancer<sup>1</sup>.

LN mapping for FIGO Clinical Stage I cervical cancer will be performed according to the NCCN Guidelines for Cervical Neoplasms, Surgical/SLN Mapping Algorithm for Early-Stage Cervical Cancer <sup>2</sup>.

In order to minimize the spillage of blue dye or IC2000 interfering with the mapping procedure when LNs are excised, mapping will be performed on one side of the pelvis


followed by the other side of the pelvis, and LN mapping with both Blue dye and PINPOINT will be completed prior to the excision of any LNs.

According to the randomization assignment, subjects randomized into the B-P Arm will be administered Blue dye first followed by the administration of IC2000. Blue dye and IC2000 will be prepared in separate syringes and administered into the cervix at the three and nine o'clock position with a superficial and deep injection. Subjects in the B-P Arm, will undergo LN mapping with Blue dye first followed by mapping with PINPOINT. LN mapping with Blue dye will be performed until the investigator identifies all blue nodes or determines that blue nodes cannot be identified. Once complete, the Investigator will begin mapping with PINPOINT until all IC2000' nodes are identified or the investigator determines that 'IC2000' nodes cannot be identified. Once mapping with both Blue dye and PINPOINT have been completed and documented, all LNs identified with Blue dye or PINPOINT will be excised.

Subjects randomized into the P-B Arm will be administered IC2000 first followed by the administration of Blue dye. Similar to the B-P Arm, IC2000 and Blue dye will be prepared in separate syringes and administered into the cervix at the three and nine o'clock position with a superficial and deep injection. Subjects in the P-B Arm, will undergo LN mapping with PINPOINT first followed by mapping with Blue dye. LN mapping will be performed until the investigator identifies all 'IC2000' nodes or determines that 'IC2000' nodes cannot be identified. Once complete, the Investigator will begin mapping with Blue dye until all 'blue' nodes are identified or the investigator determines that 'blue' nodes cannot be identified. Once mapping with both Blue dye and PINPOINT have been completed and documented, all LNs identified with Blue dye or PINPOINT will be excised.

.

The Investigator will identify 'Blue' nodes and 'IC2000' nodes based on direct visualization with white light for Blue dye and PINPOINT for IC2000 according to <u>Section 8.3.1.3</u> and <u>8.3.1.4</u> respectively. All nodes identified during the mapping procedure will be classified according to Section <u>8.3.1.5</u> and recorded in the operative CRFs.

## 8.3.1.1 Imaging Agent Dosing and Administration of Blue dye

The Blue dye solution will be prepared and administered by the appropriate qualified study and/or operating room personnel according to the method of Abu Rustum<sup>4</sup>. The cervix will be injected with Blue dye while the subject is under anesthesia in the operating room, approximately 15 minutes prior to planned mapping.

- One vial of Isosulfan Blue (1% solution) will be utilized A 22G spinal needle will be used to inject Blue dye at the 3 and 9 o'clock positions.
- At each position, a superficial (1-3 mm) and a deep (1-3 cm) injection of 1 mL of Blue dye will be made into the cervical submucosa and stroma. Blue dye should be injected at a rate of 5 to 10 seconds per injection.
- Total dose of Isosulfan blue administered will be 40 mg (10 mg/ml Isosulfan Blue, 4 x 1 ml injections/subject)

# 8.3.1.2 Imaging Agent Dosing and Administration of IC2000

Similar to administration of Blue dye solution, the IC2000 solution will be prepared and administered by the appropriate qualified study and/or operating room personnel according to



the method of Abu Rustum<sup>4</sup>. The cervix will be injected with IC2000 while the subject is under anesthesia in the operating room, approximately15 minutes prior to the planned time of imaging.

- One 25 mg vial of IC2000 will be reconstituted with 20 ml sterile water for injection to yield a 1.25 mg/ml solution immediately prior to IC2000 administration.
- A 22G spinal needle will be used to inject IC2000 at the 3 and 9 o'clock positions.
- At each position, a superficial (1-3 mm) and a deep (1-3 cm) injection of 1 mL of IC2000 will be made into the cervical submucosa and stroma.
- IC2000 should be injected at a rate of 5 to 10 seconds per injection.

The total dose of IC2000 administered will be 5 mg (4 x 1 ml injections/subject).

# 8.3.1.3 Identification of Lymph Nodes with Blue Dye

Intraoperative identification of LNs with Blue dye will be based on the following criteria:

- Direct visual identification of a node stained with Blue dye.
- Visible or palpably abnormal LNs designated as palpable masses and excised regardless of visible blue dye.

Mapping will be considered complete when all nodes meeting any of the criteria above are identified, classified and documented and the surgeon has scanned the full 360-degree area within the abdominal cavity. Blue ducts should be followed in both directions in order to identify LNs to be excised.

## 8.3.1.4 Identification of Lymph Nodes with PINPOINT

Intraoperative identification of LNs with PINPOINT will be based on the following criteria:

- Direct visual identification of a node by NIR fluorescence with IC2000 using PINPOINT.
- Visibly or palpably abnormal LNs designated as palpable masses and excised regardless of visible fluorescence.

Mapping will be considered complete when all nodes meeting any of the criteria above are identified, classified and documented and the surgeon has scanned the full 360-degree area around the injection site. Fluorescent ducts should be followed in both directions in order to identify LNs to be excised. Once all 'IC2000' nodes have been identified

#### 8.3.1.5 Classification of Lymph Nodes

All LNs identified will be classified as:

- 1. Fluorescent only
- 2. Blue only
- 3. Both (Fluorescent and blue)
- 4. Abnormal or palpably hard
- 5. Non-stained node found at termination of fluorescent duct
- 6. Non-stained node found at termination of blue duct
- 7. Non-stained node found at termination of fluorescent and blue duct

All LN identified and subsequently removed will be histologically examined to confirm the presence of lymphoid tissue according to section 8.5.



# 8.3.1.4.1 National Comprehensive Cancer Network Guidelines

The LN mapping procedure for subjects with uterine neoplasms will be performed according to the guidelines from the *NCCN* for *Uterine Neoplasms*, *SLN Algorithm for Surgical staging of Endometrial Cancer*<sup>1</sup> (Figure 2) in addition to the removal of other LNs according to standard of care.

FIGURE 2. SLN Algorithm for Surgical Staging of Endometrial Cancer



The LN mapping procedure for subjects with cervical neoplasms will be performed according to the guidelines from the NCCN for Cervical Neoplasms, Surgical/SLN Mapping Algorithm for Early-stage Cervical Cancer<sup>2</sup> (Figure 3) in addition to the removal of other LNs according to standard of care.

Novadag - CONFIDENTIAL



FIGURE 3. SLN Algorithm for Surgical Staging of Cervical Cancer



# 8.4 Post-operative Follow-up Visits (Day of discharge to Day 30)

Subjects will have standard of care assessments throughout the study according to the hospital/institution's standard procedures as well as study specific visits on the date of discharge and Day 30 (±7 days). Day 30 visit will be a telephone call and subjects will be assessed for the following throughout the study:

- Concomitant medications and procedures as described in section 6.3
- Adverse events and adverse device effects according to section 9

Although the subject may be seen by various individuals post-surgery, the study-specific visits must be conducted by a surgeon who is part of the study and has signed the Signature and Delegation Log. Any adverse events/adverse device effects, complications and outcomes of the study that occur between visits will be documented at the next study required visit.

# 8.5 Histopathology of Excised LN

The presence of lymphoid tissue for each excised LN will be confirmed by tissue analysis. All LNs will be routinely sectioned and stained with hematoxylin and eosin (H&E). LN ultra-staging will be performed according to the method of Kim et al.<sup>34</sup>. Briefly, two adjacent 5-µm sections will be cut and sectioned at each of the two levels, 50-µm apart from each paraffin block. Sections at each level will be stained with H&E and with immunohistochemistry using anticytokeratin AE1:AE3. Image Acquisition and Transmission

Videos of the image sequences acquired using PINPOINT will be recorded to a medical grade video recorder. All required images will be provided to the Sponsor by the Investigative Center.



Image files will be identified using the subject number and initials only (no information identifying the subject shall be included in the files).

## 9 EVALUATION, RECORDING, AND REPORTING OF ADVERSE EVENTS

All untoward medical occurrences either observed by the Investigator or one of his/her medical collaborators, or reported by the subject spontaneously, or in response to the direct question below, will be reported as follows:

- All events occurring before randomization should be recorded in the source documents and will be considered part of the subject's case history.
- All adverse events occurring during the study will be recorded as adverse events on the adverse event CRF.
- Events occurring as a result of the surgery will be reported as adverse events related to the surgical procedure in the adverse event CRF.
- Events related to PINPOINT will be recorded as adverse device effects in the CRF.
  - Events that are not related to PINPOINT shall be recorded as adverse events.
- Events related to PINPOINT that affect a user of the device (non-subject) are recorded as technical complaints.
- Events related to IC2000 and/or Blue dye will be recorded as adverse events related to IC2000 and/or blue dye in the adverse event CRF.

In an attempt to optimize consistency of AE reporting across centers, the subjects must be asked a standard question to elicit events. At each clinic or telephone evaluation of the subject, study personnel will ask the following questions: "Have you had any problems since your last visit?"

AEs reported on the CRF will include the date of onset, severity, relationship to PINPOINT, IC2000 and/or Blue dye, relationship to surgical procedure, date of resolution (or the fact that it is ongoing or has become chronic), action taken, and whether the AE is serious or not.

#### 9.1 Definitions

# 9.1.1 Adverse Event (AE)

Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory findings) in subjects whether or not related to the investigational medical device.

- Includes events related to the IC2000 or Blue dye.
- Includes events related to procedures involved (any procedure in the clinical investigation plan).
- Postoperative nausea or vomiting occurring during the first 24 to 48 hours, and postoperative pain related to surgical procedure is not considered an adverse event.

# FILM

9.1.2 Adverse Device Effect (ADE)

Any adverse event related to the use of PINPOINT (includes all hardware components).

Includes any event that is a result of a use error or intentional misuse.

ADEs that affect subjects will be recorded as ADEs in the AE CRF. ADEs that only affect a user (non-subject) are recorded in the technical complaint form only.

#### 9.1.3 Serious Adverse Event

(SAE) Any adverse event that:

- a. Led to a death.
- b. Led to a serious deterioration in health that either:
  - i. Resulted in a life-threatening illness or injury,
  - ii. Resulted in a permanent impairment of a body structure or a body function,
  - iii. Required in-patient hospitalization or prolongation of existing hospitalization,
  - iv. Resulted in medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function.
- c. Led to fetal distress, fetal death or a congenital abnormality or birth defect.

This includes device deficiencies that might have led to a serious adverse event if suitable action had not been taken; intervention had not been made, or if circumstances had been less fortunate. These are handled as SAEs. A planned hospitalization for pre-existing condition, or a procedure required by the protocol, without a serious deterioration in heath, is not considered to be a serious adverse event.

# 9.1.4 Unanticipated Adverse Device Effect

(UADE) Any ADE that meets the following:

- By its nature, incidence, severity or outcome has not been identified in the current version of the PINPOINT risk analysis report.
- On health or safety, any life-threatening problem or death caused by, or associated with a
  device, if that effect, problem, or death was not previously identified in nature, severity, or
  degree of incidence in the application; or any other unanticipated serious problem
  associated with a device that relates to the rights, safety, or welfare of subjects.

#### 9.2 Adverse Event Descriptions

#### 9.2.1 Intensity

The intensity of AEs, including ADEs will be characterized as mild, moderate, or severe, as follows:



Mild Usually transient, requiring no special treatment, and does not interfere

with the subject's daily activities.

Moderate Introduces a low level of inconvenience or concern to the subject and may

interfere with daily activities, but is usually ameliorated by simple

therapeutic measures.

Severe Significantly interferes with a subject's usual daily activities and requires

systemic drug therapy or other treatment, if available.

9.2.2 Relationship

Suspected There is a reasonable possibility that the AE is associated with use of the

study device or treatment (IC2000 or Blue dye), such as temporal

relationship of the event to use.

Not suspected A relationship between the AE and the study device or treatment (IC2000

or Blue dye) can reasonably be ruled out based on lack of any temporal relationship of the event to use, or when the subject's underlying condition, medical history, or other therapy provide sufficient explanation

for the observed event.

# 9.3 Reporting and Evaluation of Serious Adverse Events and Unanticipated Adverse Device Effects

Any SAE or UADE occurring in this study must be reported immediately (within 24 hours of discovery) by email to the Novadaq contact listed below:

**Attention: Alicia Wilton** 

Mobile: 905-629-3822 x209

Email: Film@novadaq.com

SAEs and UADEs will be reported to the Institutional Review Board (IRB)/Ethics Committee (EC) according to the institution's policies, but within 10 days of occurrence.

The Sponsor will be responsible for reporting SAEs/UADEs to the FDA or Health Canada in accordance with federal regulatory requirements.

The Sponsor will provide documentation of reportable events to the Investigator, as specified in Section 13.1.4.

The Investigator will ensure that the subject receives appropriate medical treatment and that the subject is followed up until the SAE or UADE resolves or becomes chronic, as defined in Section 9.4.

## 9.4 Follow-up for Adverse Device Effects and Adverse Events

Throughout the study to the final study visit contact, ADEs will be followed until they resolve or become chronic. All AEs will be followed throughout the study until the Day 30 visit. All AEs



related to the PINPOINT, IC2000, Blue dye or the mapping procedures, as determined by the Investigator, will be followed until resolution or deemed chronic

At the final study visit, new AEs, as well as follow-up information for continuing AEs, will be recorded in the CRF and source document. If an SAE or UADE is unresolved at the final study visit, it will be followed by the Investigator until it resolves or becomes chronic (as judged by the Investigator). Follow-up data for such SAEs will be recorded in the source document and reported to the safety contacts. Non-serious ongoing AEs will be followed beyond the final study visit if they are related to the study procedures at the discretion of the Investigator.

# 9.5 Reporting of Technical Complaints/Device Deficiencies

#### 9.5.1 Definitions

**Device Complaint:** A quality complaint received in writing, electronically, or orally that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness, or performance of a device product. (In this definition, "effectiveness" refers to the actual function of the device, not to how the subject responds to the action of the device. Also in this definition, "device product" refers only to devices provided by the Sponsor for clinical studies and to investigational devices.)

In this definition, safety includes the safety of a subject, user, or other person associated with the use of a medical device.

**Device Deficiency:** Inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. Device deficiencies include malfunctions, use errors and inadequate labelling.

## 9.5.2 Reporting Procedures

Any technical complaint/device deficiency should be reported to the Sponsor. Technical Complaints occurring in this study must be reported immediately (within 24 hours) by fax or email to the appropriate Novadag representative or to Novadag Quality (quality@novadag.com)

Any complaint about a device must be reported regardless of whether the defect or deficiency had any effect on a subject or on study personnel.

#### 9.6 ADEs Technical Complaints/Device Deficiencies that are UADEs

Novadaq will evaluate all ADE reports and technical complaints/device deficiencies to determine if the report meets the definition of an unanticipated adverse device effect. If Novadaq determines that it does meet the definition, an investigation will be begun immediately. Novadaq will inform the Investigator of any additional reporting requirements beyond those stated in <a href="Sections 9.4">Sections 9.4</a> and <a href="9.5">9.5</a> as applicable.

Novadaq will report the UADE and the results of any investigations to the FDA and Health Canada according to the applicable regulatory guidelines. Novadaq will also report to the Investigator(s), who will submit the required reports to their IRB/ECs within 10 working days after Novadaq first received notice of the effect.

# FILM

## 10 STATISTICAL CONSIDERATIONS

# 10.1 Primary Objective

To assess the effectiveness of intraoperative PINPOINT in identification of LNs in subjects with uterine and cervical malignancies who are undergoing LN mapping.

# 10.2 Hypotheses

To assess the effectiveness of PINPOINT in the identification of LNs, a non-inferiority test will be performed using the per-protocol (PP) analysis population.

 $H_{01}$ :  $p_t \le p_c - 0.05$  $H_{11}$ :  $p_t > p_c - 0.05$ 

Here  $p_t$  and  $p_c$  represent the effectiveness of LN mapping with PINPOINT and Blue dye respectively. We define the numerator for  $p_t$  as the number of nodes identified with PINPOINT (classifications 1, 3, 5, 7 as defined in section 8.3.1.5) and confirmed as lymphoid tissue, and we define the numerator for  $p_c$  as the number of nodes identified with Blue dye (classifications 2, 3, 6, 7 as defined in section 8.3.1.5) and confirmed as lymphoid tissue. We define the denominator for both  $p_t$  and  $p_c$  as the number of nodes identified by ANY method (classifications 1-7 as defined in section 8.3.1.5). The denominator will include excised nodes confirmed as lymphoid tissue.

A non-inferiority margin of 0.05 was determined to be clinically significant based on feedback from Investigators. Within their respective groups,  $p_t$  and  $p_c$  represent the proportion of LNs identified (and confirmed to be lymphoid tissue, See Section 8.5) with PINPOINT and Blue dye respectively divided by the total number of LNs identified and excised, across all subjects.

We will repeat the analysis described above using the as-treated (AT) analysis set as a supporting analysis of the primary outcome.

As a sensitivity analysis we will also perform the non-inferiority test using the mITT analysis set. We will also perform sensitivity analyses of the primary endpoint using a best-case and a worst-case scenario. The best-case scenario will consider nodes with missing histology to be lymphoid tissue for PINPOINT and non-lymphoid tissue for Blue dye. The worst case scenario will consider nodes with missing histology to be non-lymphoid tissue for PINPOINT and lymphoid tissue for Blue dye.

# 10.3 Statistical Analysis

We will use the  $Z_{\text{O}}$  statistic described by Nam and Kwon () in formulae (6) to derive the estimates of  $p_{\text{t}}$ ,  $p_{\text{c}}$ , and the variance of the difference between these estimates to construct the 95% 2-sided confidence interval for  $p_{\text{t}}-p_{\text{c}}$  as:

$$\left( (\hat{p}_t - \hat{p}_c) - 1.96 \times \sqrt{\widehat{var}(\hat{p}_t - \hat{p}_c)} \right), (\hat{p}_t - \hat{p}_c) + 1.96 \times \sqrt{\widehat{var}(\hat{p}_t - \hat{p}_c)} \right)$$



We will perform this analysis using the PP analysis set to test the inferiority hypothesis ( $H_{01}$ ) stated above, and if the lower bound of the interval is > -0.05 we will claim non-inferiority. If and only if we reject the null ( $H_{01}$ ) hypothesis of inferiority and claim non-inferiority we will use the mITT analysis set to test the null ( $H_{02}$ ) stated below, and if the lower bound of the interval is > 0 we will claim superiority.

$$H_{02}$$
:  $p_t = p_c$   
 $H_{12}$ :  $p_t > p_c$ 

We will repeat the analysis described above using the as-treated (AT) analysis set as a supporting analysis of the primary outcome.

As a sensitivity analysis we will also perform the non-inferiority test using the mITT analysis set. We will also perform sensitivity analyses of the primary endpoint using a best-case and a worst-case scenario. The best-case scenario will consider nodes with missing histology to be lymphoid tissue for PINPOINT and non-lymphoid tissue for Blue dye. The worst case scenario will consider nodes with missing histology to be non-lymphoid tissue for PINPOINT and lymphoid tissue for Blue dye.

# 10.4 Sample Size Considerations

The clinical literature provides an estimate of the expected effectiveness of LN mapping with ICG and Blue Dye<sup>17–28,36</sup>. 12 studies using ICG for the purposes of LN mapping have been published<sup>17–28</sup> (Table 1). Detection rates for LN mapping with ICG and Blue dye are reported to occur in a wide range (33-100% for ICG<sup>17–28</sup> and 40-80% for Blue dye<sup>36</sup>). A number of factors play a role in the identification of LN including tumor size, familiarity with LN mapping technique (learning curve) and obesity<sup>36</sup>.

A weighted average of published LN detection rates for Blue dye and ICG (i.e., PINPOINT) in gynecological cancer suggests unilateral detection rates of 91% for ICG and 80% for Blue dye. However, we assumed LN detection rates in gynecological cancer 17-28 of 84% and 80% using ICG and Blue dye, respectively. We used a lower LN detection rate of 84% for ICG and a LN detection rate at the upper end of the range for Blue dye as a conservative approach to the sample size calculation. We also assumed a non-inferiority margin of 5%.

The power calculation was performed for a 2-level hierarchical model in which nodes are nested within subject. Power was calculated as a function of the effective sample size (ESS), which is a function of the total number of nodes excised, the number of nodes within subjects (clusters), and the intra-cluster correlation (ICC). Specifically, ESS = n / VIF, where n is the total number of nodes excised across all patients, and VIF is the variance inflation factor, calculated as VIF = 1 + (m - 1) × ICC, where m is the number of nodes per subject. Because we expect to excise 3 to 4 nodes per subject, with 150 subjects we expect to excise  $3.5 \times 150 = 525$  nodes. With 3.5 nodes per subject on average and an ICC at most 0.125 we will have VIF at most 1 +  $(2 \times 3.5 - 1) \times 0.125 = 1.75$  and an ESS at least 525 / 1.75 = 300 nodes. Note that here m is twice the number of expected nodes per subject, since nodes will be identified using 2 different methods within the same subject. We expect the ICC to be at most 0.125 based on our estimate of the ICC = 0.07 from Crane et al. 18

With an ESS of at least 300 Ns we will have at least 82% power to reject H<sub>01</sub> above and claim non-inferiority of PINPOINT with respect to Blue dye. This sample size calculation was



performed using nQuery Advisor ® 7.0 (Copyright © 1995-2007, Statistical Solutions, Saugus, MA). We will test the hypothesis using a two-sided 95% confidence interval (i.e., two-sided significance level of 0.05). We will enroll subjects and identify Ns using both Blue dye and PINPOINT as described above in section 8.3.1.5 until we have at least 525 LNs identified, regardless of the method used to identify them. We expect that we will enroll approximately 150 subjects to obtain 525 nodes (based on clinical literature suggesting an average of 3-4 Ns excised per subject 17-28).

## 10.5 Data Sets to be Analyzed

# 10.5.1 Per-protocol (PP)

The Per-Protocol (PP) analysis population includes all subjects that: [1] meet critical eligibility criteria, [2] have no significant protocol deviations; and [3] have evaluable assessment endpoints for the primary endpoint.

We believe that the PP population will be the population that will most likely demonstrate a difference between Blue dye and IC2000 with respect to their ability to identify lymph nodes, should a difference exist. Thus, since we are trying to show non-inferiority of IC2000 with respect to Blue dye, we believe that using the PP population for testing non-inferiority is the conservative approach

# 10.5.2 Modified Intent to treat (mITT)

The mITT analysis population includes all randomized subjects who received at least one injection of IC2000 or Blue dye. All subjects meeting this criterion are included in the mITT population regardless of whether or not they received the minimally invasive surgical intervention or lymphatic mapping. Subjects who have the mapping procedure aborted due to circumstances such as a higher stage cancer than initially expected will not be included in the mITT. Approximately 8% of subjects are expected to have the mapping procedure aborted.

We believe the mITT population will be the population that will most likely demonstrate no difference between the Blue dye and IC2000 with respect to their ability to identify lymph nodes, because the mITT population includes subjects who may not have received the full dose of dye, and it includes subjects who may have not received lymphatic mapping, but who may have had lymph nodes identified by gross inspection. Thus, we believe that using the mITT population for testing superiority will be the conservative approach.

# 10.5.3 As-Treated (AT)

The As-Treated (AT) analysis population includes all randomized subjects in whom the intended minimally invasive surgical procedure was performed and received at least one injection of IC2000 or Blue dye. Subjects in whom the mapping procedure with PINPOINT or Blue dye is not performed are excluded from the AT population. Subjects will be analyzed according to the LN mapping procedure performed. The AT population will be used for a secondary analysis of the primary endpoint.

## 10.5.4 Safety (S)

The safety analysis population includes all randomized subjects enrolled in the study who received at least one injection of IC2000 or Blue dye. Secondary safety endpoints, including the summary of adverse events or adverse device effects in the trial, will be analyzed using this analysis population.



# 10.6 Secondary Objectives

The planned secondary out comes are intended to support product labelling. We will use the step-down method described by Benjamini and Liu<sup>37</sup> to control the false discovery rate at 0.05 (2-sided) while testing our secondary objectives.

The first secondary outcome is the ability of PINPOINT and Blue dye to detect at least one lymph node in a subject.

Let  $q_t$  and  $q_c$  represent the proportion of subjects with a least one lymph node identified (according to <u>section</u> 8.3.1.5 and confirmed by histology) with PINPOINT and Blue dye respectively, divided by the total number of subjects where mapping was attempted. That is, the numerator for  $q_t$  is the number of subjects with at least 1 node identified with PINPOINT (classifications 1, 3, 5, 7) and confirmed as lymphoid tissue, and the numerator for  $q_c$  is the number of subjects with at least 1 node identified with Blue dye (classifications 2, 3, 6, 7) and confirmed as lymphoid tissue. The denominator of both  $q_t$  and  $q_c$  is the number of subjects where mapping was attempted.

The following hypotheses will be tested:

$$H_{03}$$
:  $q_t \le q_c - 0.05$   
 $H_{13}$ :  $q_t > q_c - 0.05$ 

To test this hypothesis we will estimate the difference  $q_t - q_c$  with a 95% two-sided confidence interval. We will perform this analysis using the PP analysis set to test the inferiority hypothesis (H<sub>03</sub>) stated above, and if the lower bound of the interval is greater than -0.05 we will claim non-inferiority. If and only if we reject the inferiority hypothesis (H<sub>03</sub>) we will use the mITT analysis set to test for superiority, and if the lower bound of the interval is greater than 0 we will claim superiority.

Another secondary outcome is the bilateral LN detection rate. Let  $b_t$  and  $b_c$  represent the proportion of subjects with at least one node identified on the right side and on the left side of the pelvis and confirmed as lymphoid tissue with PINPOINT and Blue dye, respectively. That is, the numerator for  $b_t$  is the number of subjects with at least 1 node identified with PINPOINT () on the right side of the pelvis and confirmed as lymphoid tissue and at least 1 node identified with PINPOINT on the left side of the pelvis and confirmed as lymphoid tissue. Similarly, the numerator for  $b_c$  is the number of subjects with at least 1 node identified with Blue dye (classifications 2, 3, 6, 7) on the right side of the pelvis and confirmed as lymphoid tissue and at least 1 node identified with Blue dye on the left side of the pelvis and confirmed as lymphoid tissue. The denominator of both  $b_t$  and  $b_c$  is the number of subjects where mapping was attempted.

The following hypotheses will be tested:

$$H_{04}$$
:  $b_t \le b_c - 0.05$   
 $H_{14}$ :  $b_t > b_c - 0.05$ 

To test this hypothesis we will estimate the difference  $b_t - b_c$  with a 95% two-sided confidence interval. We will perform this analysis using the PP analysis set to test the inferiority hypothesis (H04) stated above, and if the lower bound of the interval is greater than -0.05 we will claim non-inferiority. If and only if we reject the inferiority hypothesis (H<sub>04</sub>) we will use the mITT analysis



set to test for superiority, and if the lower bound of the interval is greater than 0 we will claim superiority.

A third secondary outcome is the proportion of LNs identified by following lymphatic channels (ducts). Let  $d_t$  and  $d_c$  represent the proportion of nodes identified by following a duct and confirmed as lymphoid tissue with PINPOINT and Blue dye, respectively. That is, the numerator for  $d_t$  is the number of nodes identified with PINPOINT by following a duct (classifications 5, 7) and confirmed as lymphoid tissue. Similarly, the numerator for  $d_c$  is the number nodes identified with Blue dye by following a duct (classifications 6, 7) and confirmed as lymphoid tissue. We define the denominator for both  $d_t$  and  $d_c$  as the number of nodes identified by ANY method (classifications 1-7). The denominator will include excised nodes confirmed as lymphoid tissue.

The following hypotheses will be tested:

 $H_{05}$ :  $d_t \le d_c - 0.05$  $H_{15}$ :  $d_t > d_c - 0.05$ 

To test this hypothesis we will estimate the difference  $d_t - d_c$  with a 95% two-sided confidence interval. We will estimate this confidence interval in a manner similar to that described for the primary outcome. We will perform this analysis using the PP analysis set to test the inferiority hypothesis (H05) stated above, and if the lower bound of the interval is greater than -0.05 we will claim non-inferiority. If and only if we reject the inferiority hypothesis (H<sub>05</sub>) we will use the mITT analysis set to test for superiority, and if the lower bound of the interval is greater than 0 we will claim superiority.

We will also tabulate the anatomic distribution of LNs identified by each dye.

#### 10.6.1 Demographic and Baseline Data

The demographic and baseline analysis will be done for the mITT and PP data set.

The following subject variables will be summarized: age, race, body mass index, histological type (squamous cell carcinoma, adenocarcinoma, endometrioid carcinoma etc.), previous neoadjuvant therapy, FIGO stage and type of surgical intervention. Continuous variables will be summarized as mean, standard deviation, median, minimum and maximum, and categorical variables will be summarized by counts and percentages.

# 10.6.2 Safety Variables and Analysis

Safety variables will be documented and summarized for all randomized subjects enrolled in the study who received at least one injection of IC2000 or Blue dye. Safety variables will include all adverse events (AEs) and adverse device effects (ADEs), concomitant medications, and vital signs. Safety analysis will be performed on all subjects who receive IC2000 regardless of whether LN mapping was initiated or successful.

Adverse events will be coded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE). Treatment-emergent AEs and ADEs will be summarized descriptively. The number and percentage of subjects experiencing AEs and ADEs and the total number of AEs and ADEs will be summarized by system organ class and preferred term. Associated AEs that investigators suspect are related to study treatment will also be summarized. Summary of each type of event will be prepared by severity and for all severities combined.



# 10.7 Handling of Missing Data

Reasonable efforts will be made to obtain complete data for all subjects; however, missing observations will inevitably occur due to subjects lost to follow-up or noncompliance with required assessments. The reasons for missing data will be documented and evaluated (e.g. subject is deceased, lost to follow up, missed visit, etc.). In addition, the distribution of prognostic factors between subjects with data and those without data will be examined to evaluate any potential sources of bias. Any missing observations will be described in detail and evaluated for assessment of possible bias.

A sensitivity analyses of the primary and secondary endpoints will be conducted using a bestcase and a worst-case scenario. The best-case scenario will consider nodes with missing histology as lymphoid tissue for PINPOINT and as non-lymphoid tissue for Blue dye. The worstcase scenario will consider nodes with missing histology as non-lymphoid tissue for PINPOINT and as lymphoid tissue for Blue dye.

# 10.8 Pooling of Site Data

The homogeneity of safety and effectiveness results across study sites will be examined and if no significant heterogeneity is found, the results will be pooled. The justification for pooling is that all study sites will follow one Protocol, use the same device system (PINPOINT) follow the same Instructions for Use and perform mapping in accordance with NCCN guidelines. Additionally, frequent contact and monitoring of the sites will be performed to ensure that all Study sites are evaluating participants and recording Study results in a reliable and reproducible manner. It is not anticipated that any individual Study site will dominate the Study results. Therefore, it is believed that these procedures will help to ensure that the data from these Study sites can be combined and analyzed as if generated at a single site.

#### 11 ESTIMATED DURATION OF THE STUDY

The expected study duration is approximately 1 year. The study is expected to start in 2015 and take 18 months to complete enrollment.

### 12 STUDY ETHICAL CONSIDERATIONS

# 12.1 Ethical Conduct of the Study

The study will be conducted in accordance with US 21 CFR Parts 50, 54, 56, 312 and 812 as well as ICH E6: Good Clinical Practice: Consolidated Guideline. It will be constituted in keeping with the principles of ICH E8: General Considerations for Clinical Trials and Part C, Division 5 of the Canadian Food and Drug Regulations. Any additional requirements imposed by the local Institutional Review Board/Ethics Committee/Research Ethics Board or regulatory agency will be followed as necessary.

## 12.2 Informed Consent

The informed consent forms used for the study must comply with applicable laws and regulations. An Investigator must explain the medical aspects of the study, including the nature of the study and procedure, orally and in writing, in such a manner that the subject is aware of potential benefits and risks. Other elements of the informed consent process may be delegated by the



Investigator. Subjects must be informed about all aspects of the clinical study that are necessary to make the decision to participate in the clinical trial. Subjects must be informed that participation is voluntary and that they may withdraw from the study at any time, without prejudice. Documentation of the discussion and the date of informed consent must be recorded in the source documentation. Subjects must give informed consent in writing.

The informed consent process must be conducted, and the form must be signed, before the subject undergoes any screening procedures that are performed solely for the purpose of determining eligibility for the study.

### 12.3 Institutional Review Board, Ethics Committee, or Research Ethics Board (IRB)

The protocol, protocol amendments (as specified by the IRB), and the informed consent form for the proposed study, along with any other documents required by the center's IRB must be submitted by the Investigator to the center's duly constituted IRB for review and approval. The Investigator must also ensure that the IRB reviews the progress of the study on a regular basis and, if necessary, renews its approval of the study on an annual basis. A copy of each IRB approval letter must be forwarded to the Sponsor before the study is implemented. Documentation of subsequent reviews of the study must also be forwarded to the Sponsor.

# 12.4 Data and Safety Monitoring Board

The study will be reviewed annually by an independent Data and Safety Monitoring Board (DSMB). The independent statistician will prepare a report for the DSMB in advance of the scheduled review meeting using the report template provided by the DSMB. The independent statistician will also prepare a safety report for the study Principal Investigator (PI) in preparation of the DSMB meeting to review the study. A DSMB charter will outline specific safety and data monitoring procedures.

#### 13 ADMINISTRATIVE PROCEDURES

## 13.1 Sponsor's Responsibilities

#### 13.1.1 Public Disclosure of Clinical Trials

The Sponsor will submit information about this protocol to the appropriate web-based national clinical trial registry and results database in each applicable regulatory region where the study is conducted. This includes but is not limited to US National Institute of Health (<a href="https://www.clinicaltrials.gov">www.clinicaltrials.gov</a>).

# 13.1.2 Study Supplies

The Sponsor will provide the PINPOINT Endoscopic Fluorescence Imaging System along with sufficient quantities of PINPOINT LN Mapping Kits and sufficient quantities of Blue dye (Isosulfan blue).

## 13.1.3 Investigator Training

#### 13.1.3.1 Study Initiation Visit



Study centers will have a study initiation meeting to ensure the research personnel understand the protocol, study requirements, and data capture processes. This training will take place prior to enrollment of the first subject at each study center.

# 13.1.3.2 PINPOINT System

Appropriate personnel at the study centers shall be required to participate in training on the procedural use of PINPOINT as it relates to the conduct of this study (refer to Section 6.2.3).

# 13.1.4 Ongoing Communication of Safety Information During the Study

The Sponsor will provide the Investigator with documentation of UADEs and reportable events/effects, from all study centers, reported to regulatory authorities during the conduct of the study. The Investigator must forward this documentation to the IRB, as described in Section 9.

The Sponsor will also notify the Investigator about any other safety findings that could affect the safety of subjects, affect the conduct of the study, or alter the IRB's opinion about continuation of the study.

# 13.1.5 Study Monitoring

The conduct of the study will be monitored by representatives of the Sponsor to ensure compliance with the protocol, GCP and applicable regulations. A separate study specific Monitoring Plan will outline the monitoring procedures to be followed, the required access to source data and the extent of source verification planned.

### 13.1.6 Records Retention

The Sponsor must retain all documentation pertaining to the study according to Novadaq standard operating procedures.

## 13.2 Investigator's Responsibilities

#### 13.2.1 Reporting and Recording of Study Data

Data will be captured and compiled using procedures developed by the Sponsor or their representatives. All requested study data must be recorded clearly on the CRF and other study forms as required. An explanation should be provided for all missing data. Only individuals who are identified on the Study Signature and Delegation Log may enter or correct data in the CRF. Incomplete or inconsistent data on the CRFs will result in data queries that require resolution by the Investigator.

The protocol, informed consent form, protocol amendments, safety information, and other required documents must be submitted to the IRB in a timely manner, as described in Section 12.3.

### 13.2.2 Source Documentation

The Investigator must maintain adequate and accurate source documents upon which CRFs for each subject are based. They are to be separate and distinct from CRFs, except for cases in



which the Sponsor has predetermined that direct data entry into specified pages of the subject's CRF is appropriate. These records should include detailed notes on:

- The oral and written communication with the subject regarding the study treatment (including the risks and benefits of the study). The date of informed consent must be recorded in the source documentation.
- The subject's basic identifying information, such as demographics, that links the subject's source documents with the CRFs.
- All relevant observations and data on the condition of the subject throughout the study.
- The subject's exposure to PINPOINT.
- All adverse events.

# 13.2.3 Study Devices and Imaging Agents

The Investigator is responsible for ensuring the PINPOINT system, including imaging agent, and Blue dye are controlled and are used or dispensed only to subjects enrolled in the study. Only Investigators identified on the Signature and Delegation Log may use PINPOINT for the purposes of this study.

The Investigator shall keep records documenting the receipt, use, return and disposal of the study device, drugs and components.

The Investigator will ensure that PINPOINT is returned and that any other study material will be returned to the Sponsor or disposed of according to the Sponsor's instructions on completion of the study.

#### 13.2.4 Records Retention

The Investigator must ensure that clinical study records are retained according to national regulations, as documented in the clinical trial agreement entered into with the Sponsor in connection with this study.

Subject files and other source data must be kept for the maximum period of time permitted by the hospital, institution, or private practice. The Investigator must inform the Sponsor immediately if any documents are to be destroyed, to be transferred to a different facility, or to be transferred to a different owner.

## 14 DATA MANAGEMENT

Study data will be collected using paper and/or or electronic case report forms (CRFs). Data will be entered into a study specific database in one of two ways or a combination of the following:

- Center research personnel will enter study data directly into an electronic case report form which functions as an electronic data capture screen for the study database.
- Center research personnel will enter study data onto paper CRFs, which will be submitted to the Sponsor or assigned designee.

The Sponsor or designee will follow standardized procedures for data review, database cleaning and issuing/resolving queries. Procedures for data verification, validation, security and data



retention will be followed in order that the study data reported are complete, accurate and consistent with source data.

For the purpose of data analysis and presentation, the data of the original data set may be manipulated and additional variables calculated when necessary. Once the study data are completely entered, reviewed and checked, the study database will be locked and no further changes will be made.

The electronic CRFs will be created and managed using REDCap<sup>33</sup> (Research Electronic Data Capture) electronic data capture tools hosted at M.D. Anderson. REDCap (<a href="www.project-redcap.org">www.project-redcap.org</a>) is a secure, web-based application with controlled access designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless downloads to common statistical packages; and 4) procedures for importing data from external sources. In the case of multi-center studies REDCap uses Data Access Groups (DAGs) to ensure that personnel at each institution are blinded to the data from other institutions. REDCap (<a href="https://redcap.mdanderson.org">https://redcap.mdanderson.org</a>) is hosted on a secure server by M.D. Anderson Cancer Center's Department of Research Information Systems & Technology Services. REDCap has undergone a Governance Risk & Compliance Assessment (May 2014) by M.D. Anderson's Information Security Office and found to be compliant with HIPAA, Texas Administrative Codes 202-203, University of Texas Policy 165, federal regulations outlined in 21CFR Part 11, and UTMDACC Institutional Policy #ADM0335.

Those having access to the data include the study PI and research team personnel. Users are authenticated against M.D. Anderson's Active Directory system. External collaborators are given access to the database once approved by the PI, with their access expiring in 6 months but renewable in 6 months increments at the request of the PI. The application is accessed through Secure Socket Layer (SSL). All protected health information (PHI) will be removed from the data when it is exported from REDCap for analysis. All dates for a given subject will be shifted by a randomly generated number between 0 and 364, thus preserving the distance between dates. Dates for each subject will be shifted by a different randomly generated number.

Following publication study data will be archived in REDCap. Since study data may be useful for future research studies performed under separate IRB approved protocols, study data will be archived indefinitely by the sponsor. Since REDCap is a secure electronic database with controlled access, and because subject identifiers may be needed to link study data to data from



other sources under future IRB approved protocols, subject identifying information will be retained in the archived database.

# 15 POLICY FOR PUBLICATION AND PRESENTATION OF DATA

The results of the study will be published by the study group. In addition to the principal investigators, any additional authors listed separately on the manuscript will be selected based on scientific input on the design of the study, interpretation of results and on enrollment numbers. The final number of authors will depend on the journal's publication guidelines. All participating centers will be acknowledged in the main study manuscript.

The Sponsor also encourages the scientific publication of data from clinical research studies. However, Investigators may not present or publish partial or complete study results individually without participation of the study Principal Investigator as well as the Sponsor. The Principal Investigators and the Sponsor may propose appropriate scientific manuscripts or abstracts from the study data. All proposed publications must be reviewed and commented on by the Sponsor before submission for publication. The detailed procedures for the review of publications are set out in the clinical trial agreement entered into with the Sponsor in connection with this study. These procedures are in place to ensure coordination of study data publication and adequate review of data for publication against the validated study database for accuracy. Names of all Investigators and Sponsor representatives responsible for designing the study and analyzing the results will be included in the publication(s).



#### **16 REFERENCES**

- 1. The National Comprehensive Cancer Network. Uterine Neoplasms. (2015).
- 2. The National Comprehensive Cancer Network. Cervical Neoplasms. (2015).
- 3. Nam J-M and Kwon D. Non-inferiority tests for clustered matched-pair data. Statistics in Medicine. **28**, 1668-1679 (2009).
- 4. Abu-Rustum, N. R. Sentinel lymph node mapping for endometrial cancer: a modern approach to surgical staging. *J. Natl. Compr. Canc. Netw.* **12**, 288–97 (2014).
- Sentinel Lymph Node Biopsy National Cancer Institute. at <a href="http://www.cancer.gov/cancertopics/factsheet/detection/sentinel-node-biopsy">http://www.cancer.gov/cancertopics/factsheet/detection/sentinel-node-biopsy</a>
- 6. Chen, S. L., Iddings, D. M., Scheri, R. P. & Bilchik, A. J. Lymphatic Mapping and Sentinel Node Analysis: Current Concepts and Applications. *CA. Cancer J. Clin.* **56**, 292–309 (2006).
- 7. Xiong, L. *et al.* Indocyanine green fluorescence-guided sentinel node biopsy: A meta-analysis on detection rate and diagnostic performance. *Eur. J. Surg. Oncol.* **40**, 843–9 (2014).
- 8. Kamisaka, K., Yatsuji, Y., Yamada, H. & Kameda, H. The binding of indocyanine green and other organic anions to serum proteins in liver diseases. *Clin. Chim. Acta.* **53**, 255–64 (1974).
- 9. Marshall, M. V *et al.* Near-Infrared Fluorescence Imaging in Humans with Indocyanine Green: A Review and Update. *Open Surg. Oncol. J.* **2**, 12–25 (2010).
- 10. What are the key statistics about endometrial cancer? at <a href="http://www.cancer.org/cancer/endometrialcancer/detailedguide/endometrial-uterine-cancer-key-statistics">http://www.cancer.org/cancer/endometrialcancer/detailedguide/endometrial-uterine-cancer-key-statistics</a>
- 11. Canadian Cancer Statistics publication Canadian Cancer Society. at <a href="http://www.cancer.ca/en/cancer-information/cancer-101/canadian-cancer-statistics-publication/?region=pe">http://www.cancer.ca/en/cancer-information/cancer-101/canadian-cancer-statistics-publication/?region=pe</a>
- 12. What are the key statistics about cervical cancer? at <a href="http://www.cancer.org/cancer/cervicalcancer/detailedguide/cervical-cancer-key-statistics">http://www.cancer.org/cancer/cervicalcancer/detailedguide/cervical-cancer-key-statistics</a>
- 13. Koh, W.-J. *et al.* Uterine Neoplasms, Version 1.2014. *J Natl Compr Canc Netw* **12,** 248–280 (2014).
- 14. IC-GREEN (indocyanine green for injection, USP). (2012).



- 15. ICG-Pulsion (25mg/50mg powder for solution for injection) prescribing information.
- 16. PINPOINT Operator 's Manual. (USA. Rev B 2016, Rev.A, 2016).
- 17. Furukawa, N. *et al.* The usefulness of photodynamic eye for sentinel lymph node identification in patients with cervical cancer. *Tumori* **96**, 936–40 (2010).
- 18. Crane, L. M. A. *et al.* Intraoperative near-infrared fluorescence imaging for sentinel lymph node detection in vulvar cancer: first clinical results. *Gynecol. Oncol.* **120**, 291–5 (2011).
- 19. Crane, L. M. a *et al.* Intraoperative multispectral fluorescence imaging for the detection of the sentinel lymph node in cervical cancer: a novel concept. *Mol. Imaging Biol.* **13**, 1043–9 (2011).
- 20. Holloway, R. W. *et al.* Detection of sentinel lymph nodes in patients with endometrial cancer undergoing robotic-assisted staging: a comparison of colorimetric and fluorescence imaging. *Gynecol. Oncol.* **126,** 25–9 (2012).
- 21. Rossi, E. C., Ivanova, A. & Boggess, J. F. Robotically assisted fluorescence-guided lymph node mapping with ICG for gynecologic malignancies: a feasibility study. *Gynecol. Oncol.* **124**, 78–82 (2012).
- 22. Schaafsma, B. E. *et al.* Randomized comparison of near-infrared fluorescence lymphatic tracers for sentinel lymph node mapping of cervical cancer. *Gynecol. Oncol.* **127**, 126–30 (2012).
- 23. Rossi, E. C., Jackson, A., Ivanova, A. & Boggess, J. F. Detection of sentinel nodes for endometrial cancer with robotic assisted fluorescence imaging: cervical versus hysteroscopic injection. *Int. J. Gynecol. Cancer* **23**, 1704–11 (2013).
- 24. Schaafsma, B. E. *et al.* Near-infrared fluorescence sentinel lymph node biopsy in vulvar cancer: a randomised comparison of lymphatic tracers. *BJOG* **120**, 758–64 (2013).
- 25. Jewell, E. L. *et al.* Detection of sentinel lymph nodes in minimally invasive surgery using indocyanine green and near-infrared fluorescence imaging for uterine and cervical malignancies. *Gynecol. Oncol.* **133**, 274–7 (2014).
- Sinno, A. K., Fader, A. N., Roche, K. L., Giuntoli, R. L. & Tanner, E. J. A Comparison of Colorimetric versus Fluorometric Sentinel Lymph Node Mapping During Robotic Surgery for Endometrial Cancer. *Gynecol. Oncol.* (2014). doi:10.1016/j.ygyno.2014.05.022
- 27. Plante, M. *et al.* Sentinel node mapping with indocyanine green and endoscopic near- infrared fluorescence imaging in endometrial cancer. A pilot study and review of the literature. *Gynecol. Oncol.* (2015). doi:10.1016/j.ygyno.2015.03.004



- 28. How, J. *et al.* Comparing indocyanine green, technetium, and blue dye for sentinel lymph node mapping in endometrial cancer. *Gynecol. Oncol.* (2015). doi:10.1016/j.ygyno.2015.04.004
- 29. Proulx, S. T. *et al.* Quantitative imaging of lymphatic function with liposomal indocyanine green. *Cancer Res.* **70**, 7053–62 (2010).
- 30. Rosenthal, E. L., Warram, J. M., Bland, K. I. & Zinn, K. R. The status of contemporary image-guided modalities in oncologic surgery. *Ann. Surg.* **261**, 46–55 (2015).
- 31. Heuveling, D. A. *et al.* Nanocolloidal albumin-IRDye 800CW: a near-infrared fluorescent tracer with optimal retention in the sentinel lymph node. *Eur. J. Nucl. Med. Mol. Imaging* **39**, 1161–8 (2012).
- 32. Chi, C. *et al.* Use of indocyanine green for detecting the sentinel lymph node in breast cancer patients: from preclinical evaluation to clinical validation. *PLoS One* **8**, e83927 (2013).
- 33. Mylan Institutional LLC. ISOSULFAN BLUE- HIGHLIGHTS OF PRESCRIBING INFORMATION. (2013).
- 34. Kim, C. H. *et al.* Pathologic ultrastaging improves micrometastasis detection in sentinel lymph nodes during endometrial cancer staging. *Int. J. Gynecol. Cancer* **23**, 964–70 (2013)
- 35. Lesaffre, E. Use and misuse of the p-value. *Bull. NYU Hosp. Jt. Dis.* **66**, 146–9 (2008).
- 36. Kadkhodayan, S. *et al.* Sentinel node biopsy for lymph nodal staging of uterine cervix cancer: A systematic review and meta-analysis of the pertinent literature. *Eur. J. Surg. Oncol.* **41**, 1–20 (2015).